CLINICAL TRIAL: NCT02349633
Title: PHASE 1/2 OPEN-LABEL STUDY OF PF-06747775 (EPIDERMAL GROWTH FACTOR RECEPTOR T790M INHIBITOR) IN PATIENTS WITH ADVANCED EPIDERMAL GROWTH FACTOR RECEPTOR MUTANT (DEL 19 OR L858R ± T790M) NON-SMALL CELL LUNG CANCER
Brief Title: Study For Patients With NSCLC EGFR Mutations (Del 19 or L858R +/- T790M)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was ended for strategic reasons and changes in the external environment.
  The safety profile and risk benefit ratio for PF-0674775 remained unchanged.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B7971001
Record Dates: First submitted 2015-01-23; First posted 2015-01-29 (Estimated); Results first posted 2021-06-10 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-05

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: EGFRm - Epidermal Growth Factor Receptor Mutation; Advanced EGFRm (del19 or L858R +/- T790M NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — palbociclib; avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1 (Experimental): Cohort 1 will be initiated (current dose 200 mg)
  Interventions: Drug: PF-06747775
- Cohort 2A (Experimental): Cohort 2A will evaluate PF-06747775 200 mg by mouth (PO) daily (QD) in combination with palbociclib continuous PO QD dosing in 21-day cycles. The starting dose (DL1) for palbociclib will be 100 mg PO daily. Dose finding will follow mTPI method with adjustments using DLT rate.
  Interventions: Drug: PF-06747775; Drug: Palbociclib
- Cohort 2B (Experimental): Cohort 2B will be initiated once the RP2D of the PF-06747775 and palbociclib combination is determined.
  Interventions: Drug: PF-06747775; Drug: Palbociclib
- Cohort 3 (Experimental): Cohort 3 combination is PF-06747775 200 mg PO QD and avelumab 10 mg/kg IV Q2W in 28-day (4-week) cycles. Dose finding will follow the mTPI design. Once RP2D of PF-06747775 in combination with avelumab is determined, the Dose Expansion Phase will be opened.
  Interventions: Drug: PF-06747775; Drug: Avelumab

INTERVENTIONS:
Drug: PF-06747775
Drug: Palbociclib
  Arms: Cohort 2A; Cohort 2B
Drug: Avelumab
  Arms: Cohort 3

SUMMARY:
This is a Phase 1/2 study of PF-06747775 as a single agent and in combination with other cancer treatments in patients with advanced EGFRm NSCLC. The overall clinical study consists of a Phase 1 single agent dose-escalation and expansion part to determine the RP2D of PF-06747775 single agent in patients with previously-treated EGFRm NSCLC followed by sequential evaluations of PF-06747775 at the RP2D in 3 different clinical scenarios as detailed below:

* Cohort 1: Phase 2 evaluation of PF-06747775 as a single agent in previously untreated patients with advanced EGFRm NSCLC,
* Cohort 2: Phase 1b single arm evaluation of PF-06747775 in combination with palbociclib (Cohort 2A) followed by Phase 2 randomized evaluation of PF 06747775 in combination with palbociclib vs PF-06747775 single agent (Cohort 2B) in previously-treated patients with EGFRm NSCLC with a secondary T790M mutation (del 19 and T790M or L858R and T790M), and
* Cohort 3: Phase 1b evaluation of PF-06747775 in combination with avelumab in previously-treated patients with EGFRm NSCLC with a secondary T790M mutation (del 19 and T790M or L858R and T790M).

DETAILED DESCRIPTION:
There remains an unmet medical need to develop EGFR TKI agents that effectively target both the single activating mutations of del 19 and L858R, and the secondary resistance mutation T790M, while sparing WT EGFR. Drugs active against the resistance mutation will enable molecularly targeted therapy with a more favorable toxicity profile than the current standard of cytotoxic chemotherapy platinum based doublets. Furthermore, by having a wide margin of selectivity favoring the EGFR mutants versus WT EGFR, PF 06747775 is likely to be positioned to improve patient outcomes from an efficacy and safety perspective.

ELIGIBILITY:
Partial Inclusion criteria:

Evidence of histologically or cytologically confirmed diagnosis of locally advanced or metastatic EGFRm (del 19 or L858R) NSCLC:

1. As detected by local EGFR mutation test that includes QIAGEN therascreen EGFR RGQ PCR kit, Roche cobas® EGFR Mutation Test or a sponsor-approved laboratory developed test that is validated in a CLIA laboratory (with tissue submitted for central laboratory confirmation via FDA approved QIAGEN therascreen RCQ PCR kit).
2. T790M disease as follows:

   Phase 1 If a repeat biopsy was performed on the tumor following prior EGFR TKI therapy, then T790M positive disease must be present. Patients of unknown T790M status following EGFR TKI progression (ie, no post EGFR TKI progression biopsy was performed) are eligible.

   In the PK sub-studies involving food/antacid and CYP3A4 effects, patients with EGFRm (del 19 or L858R) with any T790M status are eligible to enroll.

   Studies at RP2D Cohort 1: Patients may have de novo T790M mutation, but it is not required. Cohort 2 and Cohort 3: Patients must have EGRFm (del 19 AND T790M or L858R AND T790M) NSCLC tumors as detected by local EGFR mutation test that includes QIAGEN Therascreen EGFR RGQ PCR kit, Roche cobas® EGFR Mutation Test or a sponsor-approved laboratory developed test that is validated in a CLIA laboratory, which will then be retrospectively confirmed by the central validated Thermo Fisher Scientific Oncomine Next Generation Sequencing (NGS) cancer panel test. Patients will also be enrolled if they solely test positive for EGFR (del 19 AND T790M or L858R AND T790M) NSCLC in plasma detected by local EGFR mutation test that includes QIAGEN Therascreen EGFR Plasma RGQ kit, Roche cobas® EGFR mutation test v2 (US-IVD) or Sysmex Inostic's OncoBEAMTM EGFR test or a sponsor-approved laboratory developed test that is validated in a CLIA laboratory, which will then be retrospectively confirmed by a validated cfDNA test as determined by the Sponsor.
3. Prior treatment for EGFRm NSCLC as follows:

Phase 1 Has progressed after at least 1 prior line of therapy including and EGFR TKI. Patients may have also received other lines of therapy before or after the EGFR TKI.

Studies at RP2D Cohort 1: no prior treatment for locally advanced or metastatic EGFRm NSCLC. Cohorts 2 and 3: must have had disease progression on treatment with an approved 1st or 2nd generation EGFR TKI. Patients who have been treated with a 3rd generation EGFR TKI are ineligible for this study. Patients may have had multiple lines of therapy; however, the last therapy prior to study treatment must have been an approved EGFR TKI and received within 6 weeks prior to study registration.

Patients must have at least one measurable lesion as defined by RECIST version 1.1 that has not been previously irradiated.

Tumor tissue available. Requesting formalin fixed paraffin embedded (FFPE) block or 15 unstained sections (5 micron). If a lesser amount of tissue is available, contact the sponsor. An archival specimen is acceptable for Phase 1; a de novo specimen is required for Cohorts 2, and 3 if the T790M status was confirmed by tissue biopsy.

Partial Exclusion Criteria:

For All Phases/Cohorts Previously diagnosed brain metastases, unless the patient has completed the treatment that is clinically indicated, if any, and has recovered from the acute effects of any treatment that was delivered prior to study registration, have discontinued corticosteroid treatment for these metastases prior to registration, and are neurologically stable.

Major surgery within 2 weeks prior to registration.

Radiation therapy, excluding stereotactic radiosurgery (SRS), within 1 week prior to registration.

Systemic anti cancer therapy within 2 weeks or 5 half-lives (whichever is longer) of registration excluding EGFR TKIs. Patients on EGFR TKIs must discontinue the agent for a minimum of:

* 2 days prior to registration for erlotinib or afatinib, or 3 days for gefitinib if they will be part of the lead-in single dose PF-06747775 PK study (Phase 1 Dose Escalation Single and Multiple dose PK and ECG Assessments; Phase 1 Sildenafil at MTD; and Phase 1b/2 First-Line Single Agent). Please contact the Sponsor for direction for any other EGFR TKI.
* 5 half-lives or 5 days (whichever is longer) prior to registration if they will be starting on continuous PF-06747775 dosing directly (Phase 1 PK sub-studies at RP2D; Phase 1b/2 Combination with Palbociclib; Phase 1b Combination with Avelumab).

Partial Exclusions for Cohort 2A and 2B (Palbociclib combo):

Prior treatment with a CDK 4/6 inhibitor.

Partial Exclusions for Cohort 3 (Avelumab combo):

Prior therapy with an anti PD 1, anti PD L1, anti PD L2, anti CD137, or anti cytotoxic T lymphocyte associated antigen 4 (CTLA 4) antibody (including ipilimumab, tremelimumab or any other antibody or drug specifically targeting T cell co stimulation or immune checkpoint pathways).

Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent. Patients with diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible

Use of immunosuppressive medication at time of randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2015-05-14 (Actual); Primary Completion 2020-05-28 (Actual); Study Completion 2020-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (15):
- United States (7):
  - UC San Diego Medical Center - La Jolla, La Jolla, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - Smilow Cancer Hospital at Yale-New Haven, New Haven, Connecticut
  - UPMC Cancer Pavilion, Pittsburgh, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Seattle Cancer Care Alliance, Seattle, Washington
- Australia (3):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Prince Charles Hospital, Cancer Care Services, Chermside, Queensland
- Japan (2):
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - The Cancer Institute Hospital of JFCR, Koto-ku, Tokyo
- South Korea (3):
  - Seoul National University Hospital / Department of Internal Medicine, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7971001&StudyName=Phase%201%2F2%20Open-label%20Study%20Of%20Pf-06747775%20%28epidermal%20Growth%20Factor%20Receptor%20T790m%20Inhibitor%29%20In%20Patients%20With%20Advanced%20Epidermal%20Growth%20Factor%20Receptor%20Mutant%20%28del%2019%20Or%20L858r%20%C2%B1%20T790m%29%20Non-small%20Cell%20Lung%20Cancer

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 65 participants were enrolled, assigned to study treatment and treated in the study. The study was prematurely terminated by sponsor due to an internal strategic decision and changes in the external environment. No safety concerns were related to the study termination. No enrollments occurred in Phase 1 Food Effect and Rifampin Drug-Drug Interaction (DDI) sub-study, Phase 2 Cohort 2B or Phase 1b Cohort 3 prior to study termination.
Groups:
- Phase 1 Dose-escalation: PF-06747775 25 mg QD: Participants received a single oral dose of PF-06747775 25 mg on Day -8 (+/- 3 days) in lead-in period, followed by continuous oral dosing of PF-06747775 25 mg once daily (QD) for 21-day cycles (up to a maximum of 95 weeks).
- Phase 1 Dose-escalation: PF-06747775 50 mg QD: Participants received a single oral dose of PF-06747775 50 mg on Day -8 (+/- 3 days) in lead-in period, followed by continuous oral dosing of PF-06747775 50 mg QD for 21-day cycles (up to a maximum of 72 weeks).
- Phase 1 Dose-escalation: PF-06747775 150 mg QD: Participants received a single oral dose of PF-06747775 150 mg on Day -8 (+/- 3 days) in lead-in period, followed by continuous oral dosing of PF-06747775 150 mg QD for 21-day cycles (up to a maximum of 54 weeks).
- Phase 1 Dose-escalation: PF-06747775 275 mg QD: Participants received a single oral dose of PF-06747775 275 mg on Day -8 (+/- 3 days) in lead-in period, followed by continuous oral dosing of PF-06747775 275 mg QD for 21-day cycles (up to a maximum of 128 weeks).
- Phase 1 Dose-escalation: PF-06747775 300 mg QD: Participants received a single oral dose of PF-06747775 300 mg on Day -8 (+/- 3 days) in lead-in period, followed by continuous oral dosing of PF-06747775 300 mg QD for 21-day cycles (up to a maximum of 188 weeks).
- Phase 1 Dose-escalation: PF-06747775 450 mg QD: Participants received a single oral dose of PF-06747775 450 mg on Day -8 (+/- 3 days) in lead-in period, followed by continuous oral dosing of PF-06747775 450 mg QD for 21-day cycles (up to a maximum of 195 weeks).
- Phase 1 Dose-escalation: PF-06747775 600 mg QD: Participants received a single oral dose of PF-06747775 600 mg on Day -8 (+/- 3 days) in lead-in period, followed by continuous oral dosing of PF-06747775 600 mg QD for 21-day cycles (up to a maximum of 182 weeks).
- PF-06747775 200 mg QD Group: Participants received a single oral dose of PF-06747775 200 mg on Day -4 in lead-in period, followed by continuous oral dosing of PF-06747775 200 mg QD for 21-day cycles (up to a maximum of 165 weeks). PF-06747775 200 mg QD group was a combined group of PF-06747775 200 mg QD + sildenafil 25 mg SD (Phase 1 Sildenafil sub-study), PF-06747775 200 mg QD + esomeprazole/itraconazole (Phase 1 Esomeprazole/Itraconazole sub-study), Japan Lead-in cohort (LIC) and Phase 2 Cohort 1.
- Phase 1 Sildenafil Sub-study: PF-06747775 300 mg QD + Sildenafil 25 mg SD: Participants received a single oral dose of sildenafil 25 mg on Day -8 (+/- 3 days) in lead-in period, followed by continuous oral dosing of PF-06747775 300 mg QD for 21-day cycles (up to a maximum of 121 weeks) plus a single oral dose of sildenafil 25 mg on Cycle 1 Day 11.
- Phase 1b Cohort 2A: PF-06747775 200 mg QD + Palbociclib 100 mg QD: Participants received continuous oral dosing of PF-06747775 200 mg QD plus palbociclib 100 mg QD for 21-day cycles (up to a maximum of 102 weeks).
- Phase 1 Food Effect and Rifampin DDI Sub-study: PF-06747775 + Rifampin: Participants were planned to receive continuous oral dosing of PF-06747775 at Recommended Phase 2 Dose (RP2D) QD for a 21-day cycles plus rifampin 600 mg QD through Day 10 to 21 of Cycle 1. No participants were enrolled or treated in this cohort prior to study termination.
- Phase 2 Cohort 2B: PF-06747775 + Palbociclib: Participants were planned to receive continuous oral dosing of PF-06747775 QD and palbociclib QD at RP2D for 21-day cycles. No participants were enrolled or treated in this cohort prior to study termination.
- Phase 2 Cohort 2B: PF-06747775 Single Agent: Participants were planned to received continuous oral dosing of PF-06747775 QD at RP2D for a 21-day cycles. No participants were enrolled or treated in this cohort prior to study termination.
- Phase 1b Cohort 3: PF-06747775 + Avelumab: Participants were planned to receive continuous oral dosing of PF-06747775 at RP2D QD for 28-day cycles plus intravenous dosing of avelumab 10 mg/kg every 2 weeks (Q2W) on Days 1 and 15 of each cycle. No participants were enrolled or treated in this cohort prior to study termination.
Period: Overall Study
Arm/Group | Phase 1 Dose-escalation: PF-06747775 25 mg QD | Phase 1 Dose-escalation: PF-06747775 50 mg QD | Phase 1 Dose-escalation: PF-06747775 150 mg QD | Phase 1 Dose-escalation: PF-06747775 275 mg QD | Phase 1 Dose-escalation: PF-06747775 300 mg QD | Phase 1 Dose-escalation: PF-06747775 450 mg QD | Phase 1 Dose-escalation: PF-06747775 600 mg QD | PF-06747775 200 mg QD Group | Phase 1 Sildenafil Sub-study: PF-06747775 300 mg QD + Sildenafil 25 mg SD | Phase 1b Cohort 2A: PF-06747775 200 mg QD + Palbociclib 100 mg QD | Phase 1 Food Effect and Rifampin DDI Sub-study: PF-06747775 + Rifampin | Phase 2 Cohort 2B: PF-06747775 + Palbociclib | Phase 2 Cohort 2B: PF-06747775 Single Agent | Phase 1b Cohort 3: PF-06747775 + Avelumab
Started | 4 | 3 | 4 | 4 | 3 | 4 | 4 | 29 | 5 | 5 | 0 (No participants were enrolled in this cohort/arm prior to study termination.) | 0 (No participants were enrolled in this cohort/arm prior to study termination.) | 0 (No participants were enrolled in this cohort/arm prior to study termination.) | 0 (No participants were enrolled in this cohort/arm prior to study termination.)
Completed | 4 | 2 | 4 | 2 | 1 | 3 | 3 | 13 | 3 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 1 | 0 | 2 | 2 | 1 | 1 | 16 | 2 | 5 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal of informed consent | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Transition to compassionate use | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Early termination of survival follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Termination by sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants with advanced epidermal growth factor receptor mutant (EGFRm) non-small cell lung cancer (NSCLC) were enrolled in this study. The safety analysis set included all enrolled patients who received at least 1 dose of study treatment. No enrollments occurred in Phase 1 Food Effect and Rifampin DDI sub-study, Phase 2 Cohort 2B or Phase 1b Cohort 3 prior to study termination.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 Dose-escalation: PF-06747775 25 mg QD | Phase 1 Dose-escalation: PF-06747775 50 mg QD | Phase 1 Dose-escalation: PF-06747775 150 mg QD | Phase 1 Dose-escalation: PF-06747775 275 mg QD | Phase 1 Dose-escalation: PF-06747775 300 mg QD | Phase 1 Dose-escalation: PF-06747775 450 mg QD | Phase 1 Dose-escalation: PF-06747775 600 mg QD | PF-06747775 200 mg QD Group | Phase 1 Sildenafil Sub-study: PF-06747775 300 mg QD + Sildenafil 25 mg SD | Phase 1b Cohort 2A: PF-06747775 200 mg QD + Palbociclib 100 mg QD | Phase 1 Food Effect and Rifampin DDI Sub-study: PF-06747775 + Rifampin | Phase 2 Cohort 2B: PF-06747775 + Palbociclib | Phase 2 Cohort 2B: PF-06747775 Single Agent | Phase 1b Cohort 3: PF-06747775 + Avelumab | Total
Number analyzed (Participants) | 4 | 3 | 4 | 4 | 3 | 4 | 4 | 29 | 5 | 5 | 0 | 0 | 0 | 0 | 65
Age, Continuous [Mean (Full Range); unit: Years] | 70.5 [57 to 81] | 72.0 [71 to 73] | 62.0 [52 to 69] | 60.3 [55 to 64] | 55.7 [43 to 78] | 63.5 [53 to 77] | 61.0 [46 to 74] | 58.8 [37 to 76] | 63.6 [51 to 70] | 55.0 [47 to 73] |  |  |  |  | 60.8 [37 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 3 | 4 | 0 | 0 | 3 | 19 | 3 | 3 | 0 | 0 | 0 | 0 | 40
  Male | 1 | 1 | 1 | 0 | 3 | 4 | 1 | 10 | 2 | 2 | 0 | 0 | 0 | 0 | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 1 | 2 | 1 | 2 | 0 | 1 | 2 | 4 | 1 | 2 | 0 | 0 | 0 | 0 | 16
  Asian | 3 | 1 | 2 | 2 | 3 | 3 | 2 | 24 | 4 | 3 | 0 | 0 | 0 | 0 | 47
  Other | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Unspecified | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Primary Diagnoses and Durations [Median (Full Range); unit: Years] — Duration was since histopathological diagnosis in (years) to first dosing day or primary diagnosis visit date.
  Years
    Adenocarcinoma | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 5.8 [5.8 to 5.8] | 3.2 [2.4 to 4.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 1.5 [1.4 to 1.5] | 0.2 [0.2 to 0.2] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] |  |  |  |  | 1.5 [0.2 to 5.8]
    Lung adenocarcinoma | 0.0 [0.0 to 0.0] | 9.3 [9.3 to 9.3] | 3.6 [3.2 to 4.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 1.2 [0.1 to 2.2] | 0.0 [0.0 to 0.0] | 0.9 [0.9 to 0.9] |  |  |  |  | 2.7 [0.1 to 9.3]
    Lung adenocarcinoma stage IV | 0.0 [0.0 to 0.0] | 3.4 [3.4 to 3.4] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] |  |  |  |  | 3.4 [3.4 to 3.4]
    Non-small cell lung cancer stage IV | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 4.6 [4.6 to 4.6] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] |  |  |  |  | 4.6 [4.6 to 4.6]
    Squamous cell carcinoma | 0.0 [0.0 to 0.0] | 0.8 [0.8 to 0.8] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] |  |  |  |  | 0.8 [0.8 to 0.8]
    Lung neoplasm malignant | 3.6 [2.1 to 10.4] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.9 [0.9 to 0.9] | 5.1 [0.7 to 12.9] | 4.9 [1.0 to 8.8] | 0.0 [0.0 to 0.0] |  |  |  |  | 3.4 [0.7 to 12.9]
    Non-small cell lung cancer | 0.7 [0.7 to 0.7] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 2.0 [1.8 to 2.2] | 1.0 [0.8 to 1.4] | 2.3 [0.8 to 3.2] | 3.4 [3.4 to 3.4] | 1.7 [0.7 to 6.8] | 2.9 [2.3 to 7.2] | 2.6 [1.6 to 2.7] |  |  |  |  | 1.8 [0.7 to 7.2]
    Adenocarcinoma metastatic | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 2.1 [2.1 to 2.1] |  |  |  |  | 2.1 [2.1 to 2.1]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs) During the First Cycle in Phase 1 Dose-escalation Cohorts, Japan LIC and Phase 1b Cohort 3, and First 2 Cycles in Phase 1b Cohort 2A
Description: DLT was defined as any of the following adverse events (AEs) occurring during the first cycle for Phase 1 dose-escalation cohorts, Japan LIC and Phase 1b Cohort 3, or the first 2 cycles for Phase 1b Cohort 2A of treatment, and considered attributable to study intervention: Grade 4 neutropenia >7 days; febrile neutropenia; Grade >=3 thrombocytopenia with bleeding; Grade 4 thrombocytopenia; Grade >=3 non-hematologic toxicities; Grade 4 rash, mucositis, or diarrhea; failure to receive at least 70% of planned doses; Grade 3 QTcF prolongation in asymptomatic participants; treatment-related AEs attributable to PF-06747775, palbociclib or both that caused palbociclib treatment delay >= 10 days or omission of at least 12 doses of the combination. Grade of AE was defined according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03.
Time Frame: 21 days for Phase 1 dose-escalation cohorts and Japan LIC; 42 days for Phase 1b Cohort 2A; 28 days for Phase 1b Cohort 3
Population: The analysis population included participants in Phase 1 dose-escalation cohorts, Japan LIC, Phase 1b Cohorts 2A and 3 who were eligible, received study treatment and who either experienced a DLT during the first cycle of PF-06747775 or the first 2 cycles of PF 06747775 plus palbociclib, or completed the DLT observation period.
Measure: Count of Participants; unit: Participants
Groups:
- Japan LIC: Japan LIC included Japan LIC RP2D cohort and Japan LIC PK cohort. Japanese participants received a single oral dose of PF-06747775 200 mg on Day -4 (Japan LIC RP2D cohort) or PF-06747775 100 mg on Day -7 (Japan LIC PK cohort) in lead-in period, followed by continuous dosing of PF-06747775 200 mg QD for 21-day cycles. (up to a maximum of 61 weeks).
Arm/Group | Phase 1 Dose-escalation: PF-06747775 25 mg QD | Phase 1 Dose-escalation: PF-06747775 50 mg QD | Phase 1 Dose-escalation: PF-06747775 150 mg QD | Phase 1 Dose-escalation: PF-06747775 275 mg QD | Phase 1 Dose-escalation: PF-06747775 300 mg QD | Phase 1 Dose-escalation: PF-06747775 450 mg QD | Phase 1 Dose-escalation: PF-06747775 600 mg QD | Japan LIC | Phase 1b Cohort 2A: PF-06747775 200 mg QD + Palbociclib 100 mg QD | Phase 1b Cohort 3: PF-06747775 + Avelumab
Number analyzed (Participants) | 4 | 3 | 4 | 4 | 3 | 4 | 4 | 6 | 5 | 0
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 |

2. Primary Outcome: Number of Participants With Confirmed Objective Response (OR) in PF-06747775 200 mg QD Group
Description: Number of participants with confirmed OR according to Response Evaluation Criteria in Solid Tumor (RECIST) v1.1. Complete response (CR) was defined as complete disappearance of all target lesions with the exception of nodal disease. Partial response (PR) was defined as Greater than or equal to 30% decrease under baseline of the sum of diameters of all target measurable lesions.
Time Frame: Baseline up to end of treatment (maximum of 165 weeks)
Population: The response analysis population included all participants who received at least one dose of study medication, had measurable disease and adequate baseline assessment, and at least 1 post baseline assessment during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06747775 200 mg QD Group
Number analyzed (Participants) | 29
Participants
  CR | 0
  PR | 11

3. Primary Outcome: Progression-free Survival (PFS) in Phase 2 Cohort 2B
Description: PFS was based on Kaplan-Meier estimates. PFS was defined as the time from Cycle 1 Day 1 to the date of the first documentation of objective progression (PD) or death due to any cause. PD was defined as 20% increase in the sum of diameters of target measurable lesions above the smallest sum observed (over baseline if no decrease in the sum is observed during therapy), with a minimum absolute increase of 5 mm.
Time Frame: Cycle 1 Day 1 up to the end of study (maximum of 5 years)
Population: as for outcome 2
Arm/Group | Phase 2 Cohort 2B: PF-06747775 + Palbociclib | Phase 2 Cohort 2B: PF-06747775 Single Agent
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Participants With Treatment-emergent AEs (TEAEs) in All Cohorts All Phases (All-causality)
Description: AE = any untoward medical occurrence in participant who received study treatment without regard to possibility of causal relationship. Grade 3 (Severe) events = unacceptable or intolerable events, significantly interrupting usual daily activity, require systemic drug therapy/other treatment. Grade 4 (Life-threatening) events caused participant to be in imminent danger of death. Grade 5 (Death) events = death related to an AE. Treatment-emergent events = between first dose of study treatment and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Baseline up to 28 days after last dose of study treatment (maximum of 199 weeks)
Population: The safety analysis population included all enrolled participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Dose-escalation: PF-06747775 25 mg QD | Phase 1 Dose-escalation: PF-06747775 50 mg QD | Phase 1 Dose-escalation: PF-06747775 150 mg QD | Phase 1 Dose-escalation: PF-06747775 275 mg QD | Phase 1 Dose-escalation: PF-06747775 300 mg QD | Phase 1 Dose-escalation: PF-06747775 450 mg QD | Phase 1 Dose-escalation: PF-06747775 600 mg QD | PF-06747775 200 mg QD Group | Phase 1 Sildenafil Sub-study: PF-06747775 300 mg QD + Sildenafil 25 mg SD | Phase 1b Cohort 2A: PF-06747775 200 mg QD + Palbociclib 100 mg QD | Phase 1 Food Effect and Rifampin DDI Sub-study: PF-06747775 + Rifampin | Phase 2 Cohort 2B: PF-06747775 + Palbociclib | Phase 2 Cohort 2B: PF-06747775 Single Agent | Phase 1b Cohort 3: PF-06747775 + Avelumab
Number analyzed (Participants) | 4 | 3 | 4 | 4 | 3 | 4 | 4 | 29 | 5 | 5 | 0 | 0 | 0 | 0
Participants
  All-causality AEs | 4 | 3 | 4 | 4 | 3 | 4 | 4 | 29 | 5 | 5 |  |  |  |
  Grade 3 or 4 AEs | 1 | 1 | 4 | 4 | 2 | 3 | 4 | 12 | 2 | 5 |  |  |  |
  Grade 5 AEs | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 |  |  |  |

5. Secondary Outcome: Number of Participants With TEAEs in All Cohorts All Phases (Treatment-related)
Description: Treatment-related AE was any untoward medical occurrence attributed to study treatment in a participant who received study treatment. Grade 3 (Severe) events = unacceptable or intolerable events, significantly interrupting usual daily activity, require systemic drug therapy/other treatment. Grade 4 (Life-threatening) events caused participant to be in imminent danger of death. Grade 5 (Death) events = death related to an AE. Treatment-emergent events = between first dose of study treatment and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. Treatment-related AEs were determined by the investigator.
Time Frame: Baseline up to 28 days after last dose of study treatment (maximum of 199 weeks)
Population: The safety analysis population included all enrolled participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Dose-escalation: PF-06747775 25 mg QD | Phase 1 Dose-escalation: PF-06747775 50 mg QD | Phase 1 Dose-escalation: PF-06747775 150 mg QD | Phase 1 Dose-escalation: PF-06747775 275 mg QD | Phase 1 Dose-escalation: PF-06747775 300 mg QD | Phase 1 Dose-escalation: PF-06747775 450 mg QD | Phase 1 Dose-escalation: PF-06747775 600 mg QD | PF-06747775 200 mg QD Group | Phase 1 Sildenafil Sub-study: PF-06747775 300 mg QD + Sildenafil 25 mg SD | Phase 1b Cohort 2A: PF-06747775 200 mg QD + Palbociclib 100 mg QD | Phase 1 Food Effect and Rifampin DDI Sub-study: PF-06747775 + Rifampin | Phase 2 Cohort 2B: PF-06747775 + Palbociclib | Phase 2 Cohort 2B: PF-06747775 Single Agent | Phase 1b Cohort 3: PF-06747775 + Avelumab
Number analyzed (Participants) | 4 | 3 | 4 | 4 | 3 | 4 | 4 | 29 | 5 | 5 | 0 | 0 | 0 | 0
Participants
  Treatment-related AEs | 2 | 2 | 4 | 4 | 3 | 4 | 4 | 29 | 4 | 5 |  |  |  |
  Grade 3 or 4 treatment-related AEs | 0 | 0 | 2 | 3 | 2 | 3 | 4 | 7 | 2 | 4 |  |  |  |
  Grade 5 treatment-related AEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |

6. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) in All Cohorts All Phases
Description: An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-related SAEs were determined by the investigator.
Time Frame: Baseline up to 28 days after last dose of study treatment (maximum of 199 weeks)
Population: The safety analysis population included all enrolled participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Dose-escalation: PF-06747775 25 mg QD | Phase 1 Dose-escalation: PF-06747775 50 mg QD | Phase 1 Dose-escalation: PF-06747775 150 mg QD | Phase 1 Dose-escalation: PF-06747775 275 mg QD | Phase 1 Dose-escalation: PF-06747775 300 mg QD | Phase 1 Dose-escalation: PF-06747775 450 mg QD | Phase 1 Dose-escalation: PF-06747775 600 mg QD | PF-06747775 200 mg QD Group | Phase 1 Sildenafil Sub-study: PF-06747775 300 mg QD + Sildenafil 25 mg SD | Phase 1b Cohort 2A: PF-06747775 200 mg QD + Palbociclib 100 mg QD | Phase 1 Food Effect and Rifampin DDI Sub-study: PF-06747775 + Rifampin | Phase 2 Cohort 2B: PF-06747775 + Palbociclib | Phase 2 Cohort 2B: PF-06747775 Single Agent | Phase 1b Cohort 3: PF-06747775 + Avelumab
Number analyzed (Participants) | 4 | 3 | 4 | 4 | 3 | 4 | 4 | 29 | 5 | 5 | 0 | 0 | 0 | 0
Participants
  All-causality SAEs | 2 | 1 | 3 | 3 | 0 | 3 | 2 | 3 | 0 | 1 |  |  |  |
  Treatment-related SAEs | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 1 | 0 | 1 |  |  |  |

7. Secondary Outcome: Number of Participants With Shifts of Laboratory Results From Grade <=2 at Baseline to Grade 3 or 4 Post-baseline in All Cohorts All Phases
Description: Laboratory values included hemoglobin, platelets, white blood cell count (WBC), absolute (abs) neutrophils, abs lymphocytes, abs monocytes, abs eosinophils, abs basophils, alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (Alk Phos), sodium, potassium, magnesium, chloride, total calcium, total bilirubin, blood urea nitrogen (BUN) or urea, creatinine, uric acid, glucose, albumin, phosphorous or phosphate, prothrombin time (PT) or international normalized ratio (INR), partial thromboplastin time (PTT), urinalysis and pregnancy test. Grades of laboratory results were defined by NCI CTCAE version 4.03. Grade 3 (Severe) events = unacceptable or intolerable events, significantly interrupting usual daily activity, require systemic drug therapy/other treatment. Grade 4 (Life-threatening) events caused participant to be in imminent danger of death.
Time Frame: Baseline up to the end of treatment (maximum of 195 weeks)
Population: The safety analysis population included all enrolled participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Dose-escalation: PF-06747775 25 mg QD | Phase 1 Dose-escalation: PF-06747775 50 mg QD | Phase 1 Dose-escalation: PF-06747775 150 mg QD | Phase 1 Dose-escalation: PF-06747775 275 mg QD | Phase 1 Dose-escalation: PF-06747775 300 mg QD | Phase 1 Dose-escalation: PF-06747775 450 mg QD | Phase 1 Dose-escalation: PF-06747775 600 mg QD | PF-06747775 200 mg QD Group | Phase 1 Sildenafil Sub-study: PF-06747775 300 mg QD + Sildenafil 25 mg SD | Phase 1b Cohort 2A: PF-06747775 200 mg QD + Palbociclib 100 mg QD | Phase 1 Food Effect and Rifampin DDI Sub-study: PF-06747775 + Rifampin | Phase 2 Cohort 2B: PF-06747775 + Palbociclib | Phase 2 Cohort 2B: PF-06747775 Single Agent | Phase 1b Cohort 3: PF-06747775 + Avelumab
Number analyzed (Participants) | 4 | 3 | 4 | 4 | 3 | 4 | 4 | 29 | 5 | 5 | 0 | 0 | 0 | 0
Participants
  Anemia (Grade 3) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 1 |  |  |  |
  Anemia (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |
  Hemoglobin increased (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |
  Hemoglobin increased (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |
  Lymphocyte count increased (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |
  Lymphocyte count increased (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |
  Lymphopenia (Grade 3) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 1 |  |  |  |
  Lymphopenia (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 |  |  |  |
  Abs neutrophils (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 |  |  |  |
  Abs neutrophils (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |
  Platelets (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |
  Platelets (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |
  WBC (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 |  |  |  |
  WBC (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |
  ALT (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 |  |  |  |
  ALT (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |
  Alk Phos (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |
  Alk Phos (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |
  AST (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 |  |  |  |
  AST (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |
  Total bilirubin (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |
  Total bilirubin (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |
  Creatinine (Grade 3) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 |  |  |  |
  Creatinine (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |
  Hypercalcemia (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |
  Hypercalcemia (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |
  Hyperglycemia (Grade 3) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 |  |  |  |
  Hyperglycemia (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |
  Hyperkalemia (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 |  |  |  |
  Hyperkalemia (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |
  Hypermagnesemia (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |
  Hypermagnesemia (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |
  Hypernatremia (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |
  Hypernatremia (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |
  Hypoalbuminemia (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |
  Hypoalbuminemia (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |
  Hypocalcemia (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |
  Hypocalcemia (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |
  Hypoglycemia (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |
  Hypoglycemia (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |
  Hypokalemia (Grade 3) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |
  Hypokalemia (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |
  Hypomagnesemia (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |
  Hypomagnesemia (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |
  Hyponatremia (Grade 3) | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 3 | 0 | 0 |  |  |  |
  Hyponatremia (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |
  Hypophosphatemia (Grade 3) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 |  |  |  |
  Hypophosphatemia (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |

8. Secondary Outcome: Number of Participants Meeting Categorical Criteria of QTcF Values When PF-06747775 Was Given as a Single Agent, and in Combination With Palbociclib and Avelumab.
Description: Number of participants meeting categorical criteria of QTcF values when PF-06747775 was given as a single agent in Phase 1 dose-escalation cohorts, PF-06747775 200 mg QD group (only participants in Phase 2 Cohort 1 and Japan LIC were eligible for QTcF within this combined group), and in combination with palbociclib and avelumab in Phase 1b/2 Cohorts 2A, 2B and 3. Criteria for categorization of QTcF were defined as: maximum values 450 - <480 msec, 480 - <500 msec and >=500 msec.
Time Frame: Baseline up to Cycle 4 Day 1 (maximum of 10 weeks)
Population: QTcF analysis population included all treated participants who had at least 1 ECG assessment undertaken pre dose and 1 post dose at steady state in triplicate.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Dose-escalation: PF-06747775 25 mg QD | Phase 1 Dose-escalation: PF-06747775 50 mg QD | Phase 1 Dose-escalation: PF-06747775 150 mg QD | Phase 1 Dose-escalation: PF-06747775 275 mg QD | Phase 1 Dose-escalation: PF-06747775 300 mg QD | Phase 1 Dose-escalation: PF-06747775 450 mg QD | Phase 1 Dose-escalation: PF-06747775 600 mg QD | PF-06747775 200 mg QD Group | Phase 1b Cohort 2A: PF-06747775 200 mg QD + Palbociclib 100 mg QD | Phase 2 Cohort 2B: PF-06747775 + Palbociclib | Phase 2 Cohort 2B: PF-06747775 Single Agent | Phase 1b Cohort 3: PF-06747775 + Avelumab
Number analyzed (Participants) | 4 | 3 | 4 | 4 | 3 | 4 | 4 | 9 | 5 | 0 | 0 | 0
Participants
  450 msec - <480 msec | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 |  |  |
  480 msec - <500 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |
  >=500 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |

9. Secondary Outcome: Number of Participants Meeting Categorical Criteria of QTcB Values When PF-06747775 Was Given as a Single Agent, and in Combination With Palbociclib and Avelumab.
Description: Number of participants meeting categorical criteria of QTcB values when PF-06747775 was given as a single agent in Phase 1 dose-escalation cohorts, PF-06747775 200 mg QD group (only participants in Phase 2 Cohort 1 and Japan LIC were eligible for QTcB within this combined group), and in combination with palbociclib and avelumab in Phase 1b/2 Cohorts 2A, 2B and 3. Criteria for categorization of QTcB were defined as: maximum values 450 - <480 msec, 480 - <500 msec and >=500 msec.
Time Frame: Baseline up to Cycle 4 Day 1 (maximum of 10 weeks)
Population: QTcB analysis population included all treated participants who had at least 1 ECG assessment undertaken pre dose and 1 post dose at steady state in triplicate.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Dose-escalation: PF-06747775 25 mg QD | Phase 1 Dose-escalation: PF-06747775 50 mg QD | Phase 1 Dose-escalation: PF-06747775 150 mg QD | Phase 1 Dose-escalation: PF-06747775 275 mg QD | Phase 1 Dose-escalation: PF-06747775 300 mg QD | Phase 1 Dose-escalation: PF-06747775 450 mg QD | Phase 1 Dose-escalation: PF-06747775 600 mg QD | PF-06747775 200 mg QD Group | Phase 1b Cohort 2A: PF-06747775 200 mg QD + Palbociclib 100 mg QD | Phase 2 Cohort 2B: PF-06747775 + Palbociclib | Phase 2 Cohort 2B: PF-06747775 Single Agent | Phase 1b Cohort 3: PF-06747775 + Avelumab
Number analyzed (Participants) | 4 | 3 | 4 | 4 | 3 | 4 | 4 | 9 | 5 | 0 | 0 | 0
Participants
  450 msec - <480 msec | 1 | 2 | 2 | 1 | 1 | 0 | 0 | 2 | 1 |  |  |
  480 msec - <500 msec | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 |  |  |
  >=500 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |

10. Secondary Outcome: Number of Participants With Confirmed and Unconfirmed OR in Phase 1 Cohorts
Description: Number of participants in Phase 1 cohorts with confirmed and unconfirmed OR according to RECIST v1.1. CR was defined as complete disappearance of all target lesions with the exception of nodal disease. PR was defined as Greater than or equal to 30% decrease under baseline of the sum of diameters of all target measurable lesions. Stable was defined as not qualifying for CR, PR or PD. PD was defined as 20% increase in the sum of diameters of target measurable lesions above the smallest sum observed (over baseline if no decrease in the sum is observed during therapy), with a minimum absolute increase of 5 mm. Indeterminate was defined as progression not documented.
Time Frame: Baseline up to end of treatment (maximum of 195 weeks)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Dose-escalation: PF-06747775 25 mg QD | Phase 1 Dose-escalation: PF-06747775 50 mg QD | Phase 1 Dose-escalation: PF-06747775 150 mg QD | Phase 1 Dose-escalation: PF-06747775 275 mg QD | Phase 1 Dose-escalation: PF-06747775 300 mg QD | Phase 1 Dose-escalation: PF-06747775 450 mg QD | Phase 1 Dose-escalation: PF-06747775 600 mg QD | Phase 1 Sildenafil Sub-study: PF-06747775 300 mg QD + Sildenafil 25 mg SD | Phase 1 Food Effect and Rifampin DDI Sub-study: PF-06747775 + Rifampin
Number analyzed (Participants) | 4 | 3 | 4 | 4 | 3 | 4 | 4 | 5 | 0
Participants
  CR | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  PR | 2 | 0 | 3 | 3 | 0 | 2 | 1 | 3 |
  Stable / No response | 1 | 1 | 1 | 1 | 3 | 2 | 3 | 1 |
  PD | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 |
  Indeterminate | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 |

11. Secondary Outcome: Objective Response Rate (ORR) in Phase 1b/2 Cohorts 2A, 2B and 3
Description: ORR was defined as percentage of participants with OR based assessment of CR or PR according to RECIST v1.1 that must have been confirmed ≥4 weeks later. Participants who did not have an on treatment radiographic tumor assessment due to early progression, who received anti tumor treatment other than the study medication prior to reaching a CR or PR, or who died, progressed, or dropped out for any reason prior to reaching a CR or PR were counted as non responders in the assessment of ORR. CR was defined as complete disappearance of all target lesions with the exception of nodal disease. PR was defined as Greater than or equal to 30% decrease under baseline of the sum of diameters of all target measurable lesions.
Time Frame: Baseline up to end of treatment (maximum of 108 weeks)
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 1b Cohort 2A: PF-06747775 200 mg QD + Palbociclib 100 mg QD | Phase 2 Cohort 2B: PF-06747775 + Palbociclib | Phase 2 Cohort 2B: PF-06747775 Single Agent | Phase 1b Cohort 3: PF-06747775 + Avelumab
Number analyzed (Participants) | 5 | 0 | 0 | 0
Percentage of participants | 40.0 [7.6 to 81.1] |  |  |

12. Secondary Outcome: PFS in PF-06747775 200 mg QD Group, Phase 1b Cohorts 2A and 3
Description: PFS was based on Kaplan-Meier estimates. PFS was defined as the time from Cycle 1 Day 1 to the date of the first documentation of PD or death due to any cause. PD was defined as 20% increase in the sum of diameters of target measurable lesions above the smallest sum observed (over baseline if no decrease in the sum is observed during therapy), with a minimum absolute increase of 5 mm.
Time Frame: Cycle 1 Day 1 up to the end of study (maximum of 5 years)
Population: as for outcome 2
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | PF-06747775 200 mg QD Group | Phase 1b Cohort 2A: PF-06747775 200 mg QD + Palbociclib 100 mg QD | Phase 1b Cohort 3: PF-06747775 + Avelumab
Number analyzed (Participants) | 29 | 0 | 0
Months | 8.1 [5.4 to 23.3] |  |

13. Secondary Outcome: Duration of Objective Response (DOR) in Phase 1b/2 Cohorts
Description: DOR was the time from the date of first documentation of confirmed CR or PR to the date of first documentation of PD or death due to any cause. If tumor progression data included more than 1 date, the first date was used. DOR (months) = [progression/death date - first date of OR + 1]/30.4. CR was defined as complete disappearance of all target lesions with the exception of nodal disease. PR was defined as Greater than or equal to 30% decrease under baseline of the sum of diameters of all target measurable lesions. Stable was defined as not qualifying for CR, PR or PD. PD was defined as 20% increase in the sum of diameters of target measurable lesions above the smallest sum observed (over baseline if no decrease in the sum is observed during therapy), with a minimum absolute increase of 5 mm.
Time Frame: Baseline up to the end of study (maximum of 5 years)
Population: as for outcome 2
Measure: Median (Full Range); unit: Months
Arm/Group | PF-06747775 200 mg QD Group | Phase 1b Cohort 2A: PF-06747775 200 mg QD + Palbociclib 100 mg QD | Phase 2 Cohort 2B: PF-06747775 + Palbociclib | Phase 2 Cohort 2B: PF-06747775 Single Agent | Phase 1b Cohort 3: PF-06747775 + Avelumab
Number analyzed (Participants) | 29 | 5 | 0 | 0 | 0
Months | 8.322 [2.80 to 33.59] | 11.069 [9.70 to 12.43] |  |  |

14. Secondary Outcome: Overall Survival (OS) Probability at 12 Months in Phase 1b/2 Cohorts
Description: OS probability was based on Kaplan-Meier method. OS was defined as the time from the start date to date of death due to any cause. In the absence of confirmation of death, survival time was censored at the last date the participant was known to be alive.
Time Frame: Baseline up to the end of study (maximum of 5 years)
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Groups:
- PF-06747775 200 mg QD Group: Participants received a single oral dose of PF-06747775 200 mg on Day -4 in lead-in period, followed by continuous oral dosing of PF-06747775 200 mg QD for 21-day cycles (up to a maximum of 165 weeks). PF-06747775 200 mg QD group was a combined group of PF-06747775 200 mg QD + sildenafil 25 mg SD (Phase 1 Sildenafil sub-study), PF-06747775 200 mg QD + esomeprazole/itraconazole (Phase 1 Esomeprazole/Itraconazole sub-study), Japan Lead-in cohort (LIC) and Phase 2 Cohort 1. Only participants in Japan LIC and Phase 2 Cohort 1 were eligible for OS evaluation.
Arm/Group | PF-06747775 200 mg QD Group | Phase 1b Cohort 2A: PF-06747775 200 mg QD + Palbociclib 100 mg QD | Phase 2 Cohort 2B: PF-06747775 + Palbociclib | Phase 2 Cohort 2B: PF-06747775 Single Agent | Phase 1b Cohort 3: PF-06747775 + Avelumab
Number analyzed (Participants) | 9 | 0 | 0 | 0 | 0
Percentage of participants | 87.5 [50.0 to 97.5] |  |  |  |

15. Secondary Outcome: Plasma Area Under the Curve From Zero to Infinite Time (AUCinf) of PF-06747775 as a Single Agent After Single Dose on Day -8 lead-in Period in Phase 1 Dose-escalation Cohorts and on Day -4 lead-in Period in Phase 2 Cohort 1
Description: Plasma area under the curve from zero to infinite time (AUCinf) of PF-06747775 as a single agent after single dose on Day -8 lead-in period in Phase 1 dose-escalation cohorts and on Day -4 lead-in period in Phase 2 Cohort 1. AUCinf was area under the plasma concentration versus time curve (AUC) from zero to extrapolated infinite time.
Time Frame: 1, 2, 4, 6, 8, 24, 48 and 72 hours post-dose on Day -8 (+/- 3 days) in lead-in period for Phase 1 dose-escalation cohorts and on Day -4 in lead-in period for Phase 2 Cohort 1
Population: The PK parameter analysis population included all treated participants who had sufficient information to estimate at least 1 of the PK parameters of interest for a particular analyte.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- Phase 2 Cohort 1: PF-06747775 200 mg QD: Participants received a single oral dose of PF-06747775 200 mg on Day -4 in lead-in period, followed by continuous dosing of PF-06747775 200 mg QD for 21-day cycle (up to a maximum of 28 weeks).
Arm/Group | Phase 1 Dose-escalation: PF-06747775 25 mg QD | Phase 1 Dose-escalation: PF-06747775 50 mg QD | Phase 1 Dose-escalation: PF-06747775 150 mg QD | Phase 1 Dose-escalation: PF-06747775 275 mg QD | Phase 1 Dose-escalation: PF-06747775 300 mg QD | Phase 1 Dose-escalation: PF-06747775 450 mg QD | Phase 1 Dose-escalation: PF-06747775 600 mg QD | Phase 2 Cohort 1: PF-06747775 200 mg QD
Number analyzed (Participants) | 4 | 3 | 4 | 4 | 3 | 4 | 4 | 2
ng*hr/mL | 1618 (32) | 3195 (34) | 9536 (45) | 24100 (23) | 21160 (28) | 46170 (60) | 42650 (26) | NA (NA) — Geometric mean was not reported for n<3.

16. Secondary Outcome: Maximum Concentration Observed After Dose Administration (Cmax) of PF-06747775 as a Single Agent After Single Dose on Day -8 lead-in Period in Phase 1 Dose-escalation Cohorts and on Day -4 lead-in Period in Phase 2 Cohort 1
Description: Cmax of PF-06747775 as a single agent after single dose on Day -8 lead-in period in Phase 1 dose-escalation cohorts and on Day -4 lead-in period in Phase 2 Cohort 1. Cmax was the maximum concentration after dose administration observed directly from the data.
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase 1 Dose-escalation: PF-06747775 25 mg QD | Phase 1 Dose-escalation: PF-06747775 50 mg QD | Phase 1 Dose-escalation: PF-06747775 150 mg QD | Phase 1 Dose-escalation: PF-06747775 275 mg QD | Phase 1 Dose-escalation: PF-06747775 300 mg QD | Phase 1 Dose-escalation: PF-06747775 450 mg QD | Phase 1 Dose-escalation: PF-06747775 600 mg QD | Phase 2 Cohort 1: PF-06747775 200 mg QD
Number analyzed (Participants) | 4 | 3 | 4 | 4 | 3 | 4 | 4 | 3
ng/mL | 369.3 (55) | 570.6 (14) | 2242 (29) | 3599 (13) | 3205 (19) | 5556 (27) | 6517 (12) | 2829 (132)

17. Secondary Outcome: Half-life (t1/2) of PF-06747775 as a Single Agent After Single Dose on Day -8 lead-in Period in Phase 1 Dose-escalation Cohorts and on Day -4 lead-in Period in Phase 2 Cohort 1
Description: Half-life (t1/2) of PF-06747775 as a single agent after single dose on Day -8 lead-in period in Phase 1 dose-escalation cohorts and on Day -4 lead-in period in Phase 2 Cohort 1. t1/2 was defined as the time measured for the plasma concentration to decrease by one half.
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: hrs
Arm/Group | Phase 1 Dose-escalation: PF-06747775 25 mg QD | Phase 1 Dose-escalation: PF-06747775 50 mg QD | Phase 1 Dose-escalation: PF-06747775 150 mg QD | Phase 1 Dose-escalation: PF-06747775 275 mg QD | Phase 1 Dose-escalation: PF-06747775 300 mg QD | Phase 1 Dose-escalation: PF-06747775 450 mg QD | Phase 1 Dose-escalation: PF-06747775 600 mg QD | Phase 2 Cohort 1: PF-06747775 200 mg QD
Number analyzed (Participants) | 4 | 3 | 4 | 4 | 3 | 4 | 4 | 2
hrs | 13.12 (9.615) | 12.97 (7.921) | 6.870 (1.972) | 9.907 (10.304) | 4.113 (0.611) | 9.453 (9.654) | 6.213 (3.466) | NA (NA) — Mean was not reported for n<3.

18. Secondary Outcome: Apparent Clearance (CL/F) of PF-06747775 as a Single Agent After Single Dose on Day -8 lead-in Period in Phase 1 Dose-escalation Cohorts and on Day -4 lead-in Period in Phase 2 Cohort 1
Description: Apparent clearance (CL/F) of PF-06747775 as a single agent after single dose on Day -8 lead-in period in Phase 1 dose-escalation cohorts and on Day -4 lead-in period in Phase 2 Cohort 1. CL/F was calculated as: CL/F = dose / AUCinf. AUCinf was area under the plasma concentration versus time curve (AUC) from zero to extrapolated infinite time.
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Phase 1 Dose-escalation: PF-06747775 25 mg QD | Phase 1 Dose-escalation: PF-06747775 50 mg QD | Phase 1 Dose-escalation: PF-06747775 150 mg QD | Phase 1 Dose-escalation: PF-06747775 275 mg QD | Phase 1 Dose-escalation: PF-06747775 300 mg QD | Phase 1 Dose-escalation: PF-06747775 450 mg QD | Phase 1 Dose-escalation: PF-06747775 600 mg QD | Phase 2 Cohort 1: PF-06747775 200 mg QD
Number analyzed (Participants) | 4 | 3 | 4 | 4 | 3 | 4 | 4 | 2
L/hr | 15.43 (32) | 15.64 (34) | 15.72 (45) | 11.41 (23) | 14.19 (28) | 9.756 (60) | 14.09 (25) | NA (NA) — Geometric mean was not reported for n<3.

19. Secondary Outcome: Volume of Distribution (Vz/F) of PF-06747775 as a Single Agent After Single Dose on Day -8 lead-in Period in Phase 1 Dose-escalation Cohorts and on Day -4 lead-in Period in Phase 2 Cohort 1
Description: Vz/F was defined as apparent volume of distribution. Vz/F was calculated as: Vz/F = dose / (AUCinf * kel). kel was defined as terminal phase rate constant and calculated by a linear regression of the log-linear concentration-time curve. AUCinf was area under the plasma concentration versus time curve (AUC) from zero to extrapolated infinite time.
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Phase 1 Dose-escalation: PF-06747775 25 mg QD | Phase 1 Dose-escalation: PF-06747775 50 mg QD | Phase 1 Dose-escalation: PF-06747775 150 mg QD | Phase 1 Dose-escalation: PF-06747775 275 mg QD | Phase 1 Dose-escalation: PF-06747775 300 mg QD | Phase 1 Dose-escalation: PF-06747775 450 mg QD | Phase 1 Dose-escalation: PF-06747775 600 mg QD | Phase 2 Cohort 1: PF-06747775 200 mg QD
Number analyzed (Participants) | 4 | 3 | 4 | 4 | 3 | 4 | 4 | 2
L | 248.1 (106) | 260.3 (94) | 151.0 (75) | 114.8 (103) | 83.81 (44) | 97.50 (57) | 114.8 (67) | NA (NA) — Geometric mean was not reported for n<3.

20. Secondary Outcome: Pre-dose Concentration at Steady State (Ctrough) of PF-06747775 as a Single Agent After Multiple Doses on Cycle 1 Day 11 in Phase 1 Dose-escalation Cohorts and Phase 2 Cohorts 1 and 2B
Description: Pre-dose concentration at steady state (Ctrough) of PF-06747775 as a single agent after multiple doses on Cycle 1 Day 11 in Phase 1 dose-escalation cohorts, Phase 2 Cohorts 1 and 2B. Ctrough was defined as pre-dose concentration during multiple dosing and observed directly from data.
Time Frame: Pre-dose on Cycle 1 Day 11
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase 1 Dose-escalation: PF-06747775 25 mg QD | Phase 1 Dose-escalation: PF-06747775 50 mg QD | Phase 1 Dose-escalation: PF-06747775 150 mg QD | Phase 1 Dose-escalation: PF-06747775 275 mg QD | Phase 1 Dose-escalation: PF-06747775 300 mg QD | Phase 1 Dose-escalation: PF-06747775 450 mg QD | Phase 1 Dose-escalation: PF-06747775 600 mg QD | Phase 2 Cohort 1: PF-06747775 200 mg QD | Phase 2 Cohort 2B: PF-06747775 + Palbociclib | Phase 2 Cohort 2B: PF-06747775 Single Agent
Number analyzed (Participants) | 4 | 3 | 4 | 4 | 3 | 4 | 4 | 3 | 0 | 0
ng/mL | 5.951 (83) | 15.38 (142) | 52.66 (127) | 194.55 (55) | 80.08 (64) | 283.1 (169) | 63.23 (1158) | 46.84 (302) |  |

21. Secondary Outcome: Area Under the Curve at Steady State (AUCtau) of PF-06747775 as a Single Agent After Multiple Doses on Cycle 1 Day 11 in Phase 1 Dose-escalation Cohorts and Phase 2 Cohorts 1 and 2B
Description: AUCtau was defined as area under the plasma concentration-time profile from time zero to tau, the dosing interval, where tau = 24 hours. AUCtau was calculated using Linear/Log trapezoidal method.
Time Frame: 0 (pre-dose), 1, 2, 4, 6, 8, 24 hours post-dose on Cycle 1 Day 11 for Phase 1 dose-escalation cohorts; 0 (pre-dose), 1, 2, 4, 6, 24 hours post-dose on Cycle 1 Day 11 for Phase 2 Cohorts 1 and 2B
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Phase 1 Dose-escalation: PF-06747775 25 mg QD | Phase 1 Dose-escalation: PF-06747775 50 mg QD | Phase 1 Dose-escalation: PF-06747775 150 mg QD | Phase 1 Dose-escalation: PF-06747775 275 mg QD | Phase 1 Dose-escalation: PF-06747775 300 mg QD | Phase 1 Dose-escalation: PF-06747775 450 mg QD | Phase 1 Dose-escalation: PF-06747775 600 mg QD | Phase 2 Cohort 1: PF-06747775 200 mg QD | Phase 2 Cohort 2B: PF-06747775 + Palbociclib | Phase 2 Cohort 2B: PF-06747775 Single Agent
Number analyzed (Participants) | 4 | 3 | 4 | 4 | 3 | 4 | 4 | 3 | 0 | 0
ng*hr/mL | 2067 (33) | 3605 (60) | 14830 (74) | 31490 (48) | 21500 (28) | 40770 (36) | 43060 (56) | 19990 (122) |  |

22. Secondary Outcome: CL/F of PF-06747775 as a Single Agent After Multiple Doses on Cycle 1 Day 11 in Phase 1 Dose-escalation Cohorts and Phase 2 Cohorts 1 and 2B
Description: CL/F of PF-06747775 as a single agent after multiple doses on Cycle 1 Day 11 in Phase 1 dose-escalation cohorts, Phase 2 Cohorts 1 and 2B. CL/F was calculated as: CL/F = dose / AUCtau. AUCtau was defined as area under the plasma concentration-time profile from time zero to tau, the dosing interval, where tau = 24 hours. AUCtau was calculated using Linear/Log trapezoidal method.
Time Frame: 0 (pre-dose), 1, 2, 4, 6, 8, 24 hours post-dose on Cycle 1 Day 11 for Phase 1 dose-escalation cohorts; 0 (pre-dose), 1, 2, 4, 6, 24 hours post-dose for Phase 2 Cohorts 1 and 2B
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Phase 1 Dose-escalation: PF-06747775 25 mg QD | Phase 1 Dose-escalation: PF-06747775 50 mg QD | Phase 1 Dose-escalation: PF-06747775 150 mg QD | Phase 1 Dose-escalation: PF-06747775 275 mg QD | Phase 1 Dose-escalation: PF-06747775 300 mg QD | Phase 1 Dose-escalation: PF-06747775 450 mg QD | Phase 1 Dose-escalation: PF-06747775 600 mg QD | Phase 2 Cohort 1: PF-06747775 200 mg QD | Phase 2 Cohort 2B: PF-06747775 + Palbociclib | Phase 2 Cohort 2B: PF-06747775 Single Agent
Number analyzed (Participants) | 4 | 3 | 4 | 4 | 3 | 4 | 4 | 3 | 0 | 0
L/hr | 12.11 (33) | 13.85 (60) | 10.11 (74) | 8.737 (48) | 13.92 (28) | 11.03 (35) | 12.97 (42) | 10.01 (123) |  |

23. Secondary Outcome: Observed Accumulation Ratio (Rac) of PF-06747775 as a Single Agent After Multiple Doses on Cycle 1 Day 11 in Phase 1 Dose-escalation Cohorts and Phase 2 Cohorts 1 and 2B
Description: Rac was calculated as: Rac = (steady state AUCtau) / (single dose AUC24). AUCtau was defined as area under the plasma concentration-time profile from time zero to tau, the dosing interval, where tau = 24 hours. AUCtau was calculated using Linear/Log trapezoidal method. AUC24 was defined as area under the plasma concentration-time curve from time 0 to 24 hours.
Time Frame: 1, 2, 4, 6, 8 and 24 hours post dose on Lead-in Day -8 (dose-escalation cohorts) or -4 (Cohort 1); 0 (pre-dose), 1, 2, 4, 6, 8 (except for Cohort 1) and 24 hours post dose on Cycle 1 Day 11 for dose-escalation cohorts, Cohorts 1 and 2B
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Phase 1 Dose-escalation: PF-06747775 25 mg QD | Phase 1 Dose-escalation: PF-06747775 50 mg QD | Phase 1 Dose-escalation: PF-06747775 150 mg QD | Phase 1 Dose-escalation: PF-06747775 275 mg QD | Phase 1 Dose-escalation: PF-06747775 300 mg QD | Phase 1 Dose-escalation: PF-06747775 450 mg QD | Phase 1 Dose-escalation: PF-06747775 600 mg QD | Phase 2 Cohort 1: PF-06747775 200 mg QD | Phase 2 Cohort 2B: PF-06747775 + Palbociclib | Phase 2 Cohort 2B: PF-06747775 Single Agent
Number analyzed (Participants) | 4 | 3 | 4 | 4 | 3 | 4 | 4 | 3 | 0 | 0
Ratio | 1.467 (27) | 1.202 (24) | 1.620 (40) | 1.538 (25) | 1.035 (19) | 1.108 (13) | 1.113 (16) | 1.491 (27) |  |

24. Secondary Outcome: Steady State Accumulation Ratio (Rss) of PF-06747775 as a Single Agent After Multiple Doses on Cycle 1 Day 11 in Phase 1 Dose-escalation Cohorts and Phase 2 Cohorts 1 and 2B
Description: Steady state accumulation ratio (Rss) of PF-06747775 as a single agent after multiple doses on Cycle 1 Day 11 in Phase 1 dose-escalation cohorts, Phase 2 Cohorts 1 and 2B. Rss was calculated as: Rss = (steady state AUCtau) / (single dose AUCinf). AUCtau was defined as area under the plasma concentration-time profile from time zero to tau, the dosing interval, where tau = 24 hours. AUCtau was calculated using Linear/Log trapezoidal method. AUCinf was area under the plasma concentration versus time curve (AUC) from zero to extrapolated infinite time.
Time Frame: 1, 2, 4, 6, 8, 24, 48 and 72 hours post dose on Lead-in Day -8 (dose-escalation cohorts) or Day -4 (Cohort 1); 0 (pre-dose), 1, 2, 4, 6, 8 (except for Cohort 1) and 24 hours post dose on Cycle 1 Day 11
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Phase 1 Dose-escalation: PF-06747775 25 mg QD | Phase 1 Dose-escalation: PF-06747775 50 mg QD | Phase 1 Dose-escalation: PF-06747775 150 mg QD | Phase 1 Dose-escalation: PF-06747775 275 mg QD | Phase 1 Dose-escalation: PF-06747775 300 mg QD | Phase 1 Dose-escalation: PF-06747775 450 mg QD | Phase 1 Dose-escalation: PF-06747775 600 mg QD | Phase 2 Cohort 1: PF-06747775 200 mg QD | Phase 2 Cohort 2B: PF-06747775 + Palbociclib | Phase 2 Cohort 2B: PF-06747775 Single Agent
Number analyzed (Participants) | 4 | 3 | 4 | 4 | 3 | 4 | 4 | 2 | 0 | 0
Ratio | 1.378 (28) | 1.130 (24) | 1.554 (43) | 1.576 (29) | 1.016 (19) | 1.108 (14) | 1.086 (15) | NA (NA) — Geometric mean was not reported for n<3. |  |

25. Secondary Outcome: AUCinf of Sildenafil Dosed Alone on Day -8 lead-in Period in Phase 1 Sildenafil Sub-study
Description: AUCinf of sildenafil dosed alone and in combination with PF-06747775 200 mg or 300 mg on Day -8 lead-in period in Phase 1 Sildenafil sub-study. AUCinf was defined as area under the plasma concentration versus time curve from zero to extrapolated infinite time.
Time Frame: 0.5, 1, 2, 3, 4, 6, 8 and 24 hours post-dose on Day -8 (+/- 3 days) in lead-in period
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- Phase 1 Sildenafil Sub-study: PF-06747775 200 mg QD + Sildenafil 25 mg: Participants received a single dose of sildenafil 25 mg on Day -8 (+/- 3 days) in lead-in period, followed by continuous dosing of PF-06747775 200 mg QD through Cycle 1 Day 1 to Cycle 1 Day 11 plus a single dose of sildenafil 25 mg on Cycle 1 Day 11 (up to a maximum of 165 weeks).
Arm/Group | Phase 1 Sildenafil Sub-study: PF-06747775 200 mg QD + Sildenafil 25 mg | Phase 1 Sildenafil Sub-study: PF-06747775 300 mg QD + Sildenafil 25 mg SD
Number analyzed (Participants) | 7 | 5
ng*hr/mL | 757.7 (61) | 459.1 (41)

26. Secondary Outcome: Cmax of Sildenafil Dosed Alone on Day -8 lead-in Period in Phase 1 Sildenafil Sub-study
Description: Cmax values for sildenafil were analyzed using a mixed effects model with treatment as fixed effect and participant as random effect to estimate the effect of steady state PF-06747775 on sildenafil exposure. Cmax was the maximum concentration after dose administration observed directly from the data.
Time Frame: 0.5, 1, 2, 3, 4, 6, 8 and 24 hours post dose on Day -8 (+/- 3 days) in lead-in period
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase 1 Sildenafil Sub-study: PF-06747775 200 mg QD + Sildenafil 25 mg | Phase 1 Sildenafil Sub-study: PF-06747775 300 mg QD + Sildenafil 25 mg SD
Number analyzed (Participants) | 7 | 5
ng/mL | 182.5 (80) | 148.4 (46)

27. Secondary Outcome: CL/F of Sildenafil Dosed Alone on Day -8 lead-in Period in Phase 1 Sildenafil Sub-study
Description: CL/F of sildenafil dosed alone on Day -8 lead-in period in Phase 1 Sildenafil sub-study. CL/F was calculated as: CL/F = dose / AUCinf. AUCinf was area under the plasma concentration versus time curve (AUC) from zero to extrapolated infinite time.
Time Frame: 0.5, 1, 2, 3, 4, 6, 8 and 24 hours post dose on Day -8 (+/- 3 days) in lead-in period
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Phase 1 Sildenafil Sub-study: PF-06747775 200 mg QD + Sildenafil 25 mg | Phase 1 Sildenafil Sub-study: PF-06747775 300 mg QD + Sildenafil 25 mg SD
Number analyzed (Participants) | 7 | 5
L/hr | 33.03 (61) | 54.39 (41)

28. Secondary Outcome: AUCinf of Sildenafil Dosed in Combination With PF-06747775 200 mg or 300 mg on Cycle 1 Day 11 in Phase 1 Sildenafil Sub-study
Description: as for outcome 25
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8 and 24 hours post-dose on Cycle 1 Day 11 (+/- 4 days)
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Phase 1 Sildenafil Sub-study: PF-06747775 200 mg QD + Sildenafil 25 mg | Phase 1 Sildenafil Sub-study: PF-06747775 300 mg QD + Sildenafil 25 mg SD
Number analyzed (Participants) | 6 | 5
ng*hr/mL | 429.1 (84) | 298.3 (39)

29. Secondary Outcome: Cmax of Sildenafil Dosed in Combination With PF-06747775 200 mg or 300 mg on Cycle 1 Day 11 in Phase 1 Sildenafil Sub-study
Description: Cmax values for sildenafil were analyzed using a mixed effects model with treatment as fixed effect and participant as random effect to estimate the effect of steady state PF-06747775 on sildenafil exposure.
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8 and 24 hours post-dose on Cycle 1 Day 11 (+/- 4 days)
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase 1 Sildenafil Sub-study: PF-06747775 200 mg QD + Sildenafil 25 mg | Phase 1 Sildenafil Sub-study: PF-06747775 300 mg QD + Sildenafil 25 mg SD
Number analyzed (Participants) | 6 | 5
ng/mL | 204.5 (67) | 87.57 (29)

30. Secondary Outcome: CL/F of Sildenafil Dosed in Combination With PF-06747775 200 mg or 300 mg on Cycle 1 Day 11 in Phase 1 Sildenafil Sub-study
Description: CL/F of sildenafil dosed alone and in combination with PF-06747775 200 mg or 300 mg on Day -8 lead-in period and Cycle 1 Day 11 in Phase 1 Sildenafil sub-study. CL/F was calculated as: CL/F = dose / AUCinf. AUCinf was area under the plasma concentration versus time curve (AUC) from zero to extrapolated infinite time.
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8 and 24 hours post-dose on Cycle 1 Day 11 (+/- 4 days)
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Phase 1 Sildenafil Sub-study: PF-06747775 200 mg QD + Sildenafil 25 mg | Phase 1 Sildenafil Sub-study: PF-06747775 300 mg QD + Sildenafil 25 mg SD
Number analyzed (Participants) | 6 | 5
L/hr | 58.20 (84) | 83.88 (40)

31. Secondary Outcome: AUCtau of PF-06747775 at RP2D Under Fed and Overnight Fasted Conditions in Phase 1 Food Effect and Rifampin DDI Sub-study
Description: AUCtau of PF-06747775 at the RP2D under fed and overnight fasted conditions in Phase 1 Food Effect and Rifampin DDI sub-study. AUCtau was defined as area under the plasma concentration-time profile from time zero to tau, the dosing interval, where tau = 24 hours. AUCtau was calculated using Linear/Log trapezoidal method.
Time Frame: Pre-dose, 1, 2, 4, 6, 8 and 24 hours post dose of PF-06747775 on Cycle 1 Days 8 and 9
Population: as for outcome 15
Arm/Group | Phase 1 Food Effect and Rifampin DDI Sub-study: PF-06747775 + Rifampin
Number analyzed (Participants) | 0

32. Secondary Outcome: Cmax of PF-06747775 at RP2D Under Fed and Overnight Fasted Conditions in Phase 1 Food Effect and Rifampin DDI Sub-study
Description: Cmax of PF-06747775 at the RP2D under fed and overnight fasted conditions in Phase 1 Food Effect and Rifampin DDI sub-study. Cmax was the maximum concentration after dose administration observed directly from the data.
Time Frame: Pre-dose, 1, 2, 4, 6, 8 and 24 hours post dose of PF-06747775 on Cycle 1 Days 8 and 9
Population: as for outcome 15
Arm/Group | Phase 1 Food Effect and Rifampin DDI Sub-study: PF-06747775 + Rifampin
Number analyzed (Participants) | 0

33. Secondary Outcome: AUCtau of PF-06747775 at RP2D When Dosed Alone and After Esomeprazole/Itraconazole Treatment in Phase 1 Esomeprazole-Itraconazole DDI Sub-study
Description: AUCtau of PF-06747775 at the RP2D when dosed alone and after esomeprazole/itraconazole treatment in Phase 1 Esomeprazole-Itraconazole DDI sub-study. AUCtau was defined as area under the plasma concentration-time profile from time zero to tau, the dosing interval, where tau = 24 hours. AUCtau was calculated using Linear/Log trapezoidal method.
Time Frame: 0 (pre-dose), 1, 2, 4, 6, 8 and 24 hours post dose of PF-06747775 on Cycle 1 Days 8, 13 and 21
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- Phase 1 Esomeprazole-Itraconazole DDI Sub-study: PF-06747775 200 mg + Esomeprazole/Itraconazole: Participants received PF-06747775 QD for 21-day cycle at 200 mg on Cycle 1 Day 1-14 then 100 mg starting from Cycle 1 Day 15. On Cycle 1 Day 9-13, a 40 mg dose of esomeprazole was given to participants 2 hours prior to PF-06747775. On Cycle 1 Day 17-20, a 200 mg dose of itraconazole was given to participants at the same time with PF-06747775. On Cycle 1 Day 21, itraconazole 200 mg was given to participants 3 hours prior to PF-06747775 (up to a maximum of 165 weeks).
Arm/Group | Phase 1 Esomeprazole-Itraconazole DDI Sub-study: PF-06747775 200 mg + Esomeprazole/Itraconazole
Number analyzed (Participants) | 13
ng*hr/mL
  Cycle 1 Day 8 | 17200 (45)
  Cycle 1 Day 13 | 14340 (35)
  Cycle 1 Day 21 | 10010 (54)

34. Secondary Outcome: Cmax of PF-06747775 at RP2D When Dosed Alone and After Esomeprazole/Itraconazole Treatment in Phase 1 Esomeprazole-Itraconazole DDI Sub-study
Description: Cmax of PF-06747775 at RP2D when dosed alone and after esomeprazole/itraconazole treatment in Phase 1 Esomeprazole-Itraconazole DDI sub-study. Cmax was the maximum concentration after dose administration observed directly from the data.
Time Frame: 0 (pre-dose), 1, 2, 4, 6, 8 and 24 hours post dose of PF-06747775 on Cycle 1 Days 8, 13 and 21
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase 1 Esomeprazole-Itraconazole DDI Sub-study: PF-06747775 200 mg + Esomeprazole/Itraconazole
Number analyzed (Participants) | 13
ng/mL
  Cycle 1 Day 8 | 2597 (46)
  Cycle 1 Day 13 | 2015 (37)
  Cycle 1 Day 21 | 1592 (68)

35. Secondary Outcome: AUCtau of PF-06747775 at RP2D Dosed Alone and After Rifampin Treatment in Phase 1 Food Effect and Rifampin DDI Sub-study
Description: AUCtau of PF-06747775 at RP2D dosed alone and after rifampin treatment in Phase 1 Food Effect and Rifampin DDI sub-study. AUCtau was defined as area under the plasma concentration-time profile from time zero to tau, the dosing interval, where tau = 24 hours. AUCtau was calculated using Linear/Log trapezoidal method.
Time Frame: Pre-dose, 1, 2, 4, 6, 8 and 24 hours post dose of PF-06747775 on Cycle 1 Day 21
Population: as for outcome 15
Arm/Group | Phase 1 Food Effect and Rifampin DDI Sub-study: PF-06747775 + Rifampin
Number analyzed (Participants) | 0

36. Secondary Outcome: Cmax of PF-06747775 at RP2D Dosed Alone and After Rifampin Treatment in Phase 1 Food Effect and Rifampin DDI Sub-study
Description: Cmax of PF-06747775 at RP2D dosed alone and after rifampin treatment in Phase 1 Food Effect and Rifampin DDI sub-study. Cmax was the maximum concentration after dose administration observed directly from the data.
Time Frame: Pre-dose, 1, 2, 4, 6, 8 and 24 hours post dose of PF-06747775 on Cycle 1 Day 21
Population: as for outcome 15
Arm/Group | Phase 1 Food Effect and Rifampin DDI Sub-study: PF-06747775 + Rifampin
Number analyzed (Participants) | 0

37. Secondary Outcome: AUCtau of PF-06747775 Following Multiple Doses When Given in Combination With Palbociclib on Cycle 1 Day 15 in Phase 1b Cohort 2A and Phase 2 Cohort 2B
Description: AUCtau of PF-06747775 following multiple doses when given in combination with palbociclib on Cycle 1 Day 15 in Phase 1b Cohort 2A and Phase 2 Cohort 2B. AUCtau was defined as area under the plasma concentration-time profile from time zero to tau, the dosing interval, where tau = 24 hours. AUCtau was calculated using Linear/Log trapezoidal method.
Time Frame: 0 (pre-dose), 1, 2, 4, 6 and 24 hours post dose on Cycle 1 Day 15
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Phase 1b Cohort 2A: PF-06747775 200 mg QD + Palbociclib 100 mg QD | Phase 2 Cohort 2B: PF-06747775 + Palbociclib
Number analyzed (Participants) | 4 | 0
ng*hr/mL | 17040 (91) |

38. Secondary Outcome: Cmax of PF-06747775 Following Multiple Doses When Given in Combination With Palbociclib on Cycle 1 Day 15 in Phase 1b Cohort 2A and Phase 2 Cohort 2B
Description: Cmax of PF-06747775 following multiple doses when given in combination with palbociclib on Cycle 1 Day 15 in Phase 1b Cohort 2A and Phase 2 Cohort 2B. Cmax was the maximum concentration after dose administration observed directly from the data.
Time Frame: 0 (pre-dose), 1, 2, 4, 6 and 24 hours post dose on Cycle 1 Day 15
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase 1b Cohort 2A: PF-06747775 200 mg QD + Palbociclib 100 mg QD | Phase 2 Cohort 2B: PF-06747775 + Palbociclib
Number analyzed (Participants) | 4 | 0
ng/mL | 2757 (87) |

39. Secondary Outcome: CL/F of PF-06747775 Following Multiple Doses When Given in Combination With Palbociclib on Cycle 1 Day 15 in Phase 1b Cohort 2A and Phase 2 Cohort 2B
Description: CL/F of PF-06747775 following multiple doses when given in combination with palbociclib on Cycle 1 Day 15 in Phase 1b Cohort 2A and Phase 2 Cohort 2B. CL/F was calculated as: CL/F = dose / AUCtau. AUCtau was defined as area under the plasma concentration-time profile from time zero to tau, the dosing interval, where tau = 24 hours. AUCtau was calculated using Linear/Log trapezoidal method.
Time Frame: 0 (pre-dose), 1, 2, 4, 6 and 24 hours post dose on Cycle 1 Day 15
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Phase 1b Cohort 2A: PF-06747775 200 mg QD + Palbociclib 100 mg QD | Phase 2 Cohort 2B: PF-06747775 + Palbociclib
Number analyzed (Participants) | 4 | 0
L/hr | 11.74 (91) |

40. Secondary Outcome: Ctrough of PF-06747775 Following Multiple Doses When Given in Combination With Palbociclib on Day 15 of Cycles 1-2 and Day 1 of Cycles 2-4 in Phase 1b Cohort 2A and Phase 2 Cohort 2B
Description: Ctrough of PF-06747775 following multiple doses when given in combination with palbociclib on Day 15 of Cycles 1-2 and Day 1 of Cycles 2-4 in Phase 1b Cohort 2A and Phase 2 Cohort 2B. Ctrough was defined as pre-dose concentration during multiple dosing and observed directly from data.
Time Frame: Pre-dose on Day 15 of Cycles 1-2 and Day 1 of Cycles 2-4
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase 1b Cohort 2A: PF-06747775 200 mg QD + Palbociclib 100 mg QD | Phase 2 Cohort 2B: PF-06747775 + Palbociclib
Number analyzed (Participants) | 4 | 0
ng/mL
  Cycle 1 Day 15 | 57.73 (91) |
  Cycle 2 Day 1 | 29.44 (58) |
  Cycle 2 Day 15 | 48.39 (30) |
  Cycle 3 Day 1 | 42.68 (56) |
  Cycle 4 Day 1 | 35.12 (38) |

41. Secondary Outcome: Ctrough of PF-06747775 Following Multiple Doses When Given in Combination With Avelumab on Cycle 1 Day 15 in Phase 1b Cohort 3
Description: Ctrough of PF-06747775 following multiple doses when given in combination with avelumab on Cycle 1 Day 15 in Phase 1b Cohort 3. Ctrough was defined as pre-dose concentration during multiple dosing and observed directly from data.
Time Frame: Pre-dose on Cycle 1 Day 15
Population: as for outcome 15
Arm/Group | Phase 1b Cohort 3: PF-06747775 + Avelumab
Number analyzed (Participants) | 0

42. Secondary Outcome: AUCtau of Palbociclib Following Multiple Doses When Given in Combination With PF-06747775 on Cycle 1 Day 15 in Phase 1b Cohort 2A and Phase 2 Cohort 2B
Description: AUCtau of palbociclib following multiple doses when given in combination with PF-06747775 on Cycle 1 Day 15 in Phase 1b Cohort 2A and Phase 2 Cohort 2B. AUCtau was defined as area under the plasma concentration-time profile from time zero to tau, the dosing interval, where tau = 24 hours. AUCtau was calculated using Linear/Log trapezoidal method.
Time Frame: 0 (pre-dose), 1, 2, 4, 6 and 24 hours post dose on Cycle 1 Day 15
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Phase 1b Cohort 2A: PF-06747775 200 mg QD + Palbociclib 100 mg QD | Phase 2 Cohort 2B: PF-06747775 + Palbociclib
Number analyzed (Participants) | 4 | 0
ng*hr/mL | 1420 (42) |

43. Secondary Outcome: Cmax of Palbociclib Following Multiple Doses When Given in Combination With PF-06747775 on Cycle 1 Day 15 in Phase 1b Cohort 2A and Phase 2 Cohort 2B
Description: Cmax of palbociclib following multiple doses when given in combination with PF-06747775 on Cycle 1 Day 15 in Phase 1b Cohort 2A and Phase 2 Cohort 2B. Cmax was the maximum concentration after dose administration observed directly from the data.
Time Frame: 0 (pre-dose), 1, 2, 4, 6 and 24 hours post dose on Cycle 1 Day 15
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase 1b Cohort 2A: PF-06747775 200 mg QD + Palbociclib 100 mg QD | Phase 2 Cohort 2B: PF-06747775 + Palbociclib
Number analyzed (Participants) | 4 | 0
ng/mL | 78.93 (39) |

44. Secondary Outcome: Ctrough of Palbociclib Following Multiple Doses When Given in Combination With PF-06747775 on Day 15 of Cycles 1-2 and Day 1 of Cycles 2-4 in Phase 1b Cohort 2A and Phase 2 Cohort 2B
Description: Ctrough of palbociclib following multiple doses when given in combination with PF-06747775 on Day 15 of Cycles 1-2 and Day 1 of Cycles 2-4 in Phase 1b/2 Cohorts 2A and 2B. Ctrough was defined as pre-dose concentration during multiple dosing and observed directly from data.
Time Frame: Pre-dose on Day 15 of Cycles 1-2 and Day 1 of Cycles 2-4
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase 1b Cohort 2A: PF-06747775 200 mg QD + Palbociclib 100 mg QD | Phase 2 Cohort 2B: PF-06747775 + Palbociclib
Number analyzed (Participants) | 4 | 0
ng/mL
  Cycle 1 Day 15 | 40.46 (59) |
  Cycle 2 Day 1 | 28.83 (57) |
  Cycle 2 Day 15 | 32.80 (42) |
  Cycle 3 Day 1 | 23.82 (34) |
  Cycle 4 Day 1 | 25.85 (54) |

45. Secondary Outcome: Ctrough of Avelumab When Given in Combination With PF-06747775 on Day 1 of Cycles 1-3 and Cycle 1 Day 15 in Phase 1b Cohort 3
Description: Ctrough of avelumab when given in combination with PF-06747775 on Day 1 of Cycles 1-3 and Cycle 1 Day 15 in Phase 1b Cohort 3. Ctrough was defined as pre-dose concentration during multiple dosing and observed directly from data.
Time Frame: Pre-dose on Day 1 of Cycles 1-3 and Cycle 1 Day 15
Population: as for outcome 15
Arm/Group | Phase 1b Cohort 3: PF-06747775 + Avelumab
Number analyzed (Participants) | 0

46. Secondary Outcome: Cmax of Avelumab When Given in Combination With PF-06747775 on Day 1 of Cycles 1-3 and Cycle 1 Day 15 in Phase 1b Cohort 3
Description: Cmax of avelumab when given in combination with PF-06747775 on Day 1 of Cycles 1-3 and Cycle 1 Day 15 in Phase 1b Cohort 3. Cmax was the end of infusion peak concentration observed directly from data.
Time Frame: End of infusion of avelumab on Day 1 of Cycles 1-3 and Cycle 1 Day 15
Population: as for outcome 15
Arm/Group | Phase 1b Cohort 3: PF-06747775 + Avelumab
Number analyzed (Participants) | 0

47. Secondary Outcome: Number of Participants With Epidermal Growth Factor Receptor (EGFR) Mutations in Tumor Tissue in All Cohorts All Phases
Description: Number of participants with EGFR mutations in tumor tissue in all cohorts all phases. EGFR mutation assessments in tumor tissue included the mutations statuses of exon 19 deletion (del 19), exon 21 (L858R), G719X, L861Q, S768I, exon 20 insertions and T790M.
Time Frame: Baseline
Population: The biomarker analysis set is defined as all participants in the safety analysis set who had at least one screening and post treatment biomarker assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Dose-escalation: PF-06747775 25 mg QD | Phase 1 Dose-escalation: PF-06747775 50 mg QD | Phase 1 Dose-escalation: PF-06747775 150 mg QD | Phase 1 Dose-escalation: PF-06747775 275 mg QD | Phase 1 Dose-escalation: PF-06747775 300 mg QD | Phase 1 Dose-escalation: PF-06747775 450 mg QD | Phase 1 Dose-escalation: PF-06747775 600 mg QD | PF-06747775 200 mg QD Group | Phase 1 Sildenafil Sub-study: PF-06747775 300 mg QD + Sildenafil 25 mg SD | Phase 1b Cohort 2A: PF-06747775 200 mg QD + Palbociclib 100 mg QD | Phase 1 Food Effect and Rifampin DDI Sub-study: PF-06747775 + Rifampin | Phase 2 Cohort 2B: PF-06747775 + Palbociclib | Phase 2 Cohort 2B: PF-06747775 Single Agent | Phase 1b Cohort 3: PF-06747775 + Avelumab
Number analyzed (Participants) | 4 | 3 | 4 | 4 | 3 | 4 | 4 | 29 | 5 | 5 | 0 | 0 | 0 | 0
Participants
  del 19: Negative | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 10 | 0 | 2 |  |  |  |
  del 19: Positive | 2 | 2 | 2 | 3 | 2 | 2 | 2 | 16 | 2 | 2 |  |  |  |
  del 19: Uninformative | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 0 | 0 |  |  |  |
  del 19: Not done | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 3 | 1 |  |  |  |
  L858R: Negative | 3 | 2 | 2 | 3 | 2 | 2 | 2 | 17 | 2 | 2 |  |  |  |
  L858R: Positive | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 9 | 0 | 2 |  |  |  |
  L858R: Uninformative | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 0 | 0 |  |  |  |
  L858R: Not done | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 3 | 1 |  |  |  |
  G719X: Negative | 3 | 3 | 3 | 3 | 2 | 2 | 3 | 26 | 2 | 4 |  |  |  |
  G719X: Positive | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |
  G719X: Uninformative | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 0 | 0 |  |  |  |
  G719X: Not done | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 3 | 1 |  |  |  |
  L861Q: Negative | 3 | 3 | 3 | 3 | 2 | 2 | 3 | 26 | 2 | 4 |  |  |  |
  L861Q: Positive | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |
  L861Q: Uninformative | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 0 | 0 |  |  |  |
  L861Q: Not done | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 3 | 1 |  |  |  |
  S768I: Negative | 3 | 3 | 3 | 3 | 2 | 2 | 3 | 26 | 2 | 4 |  |  |  |
  S768I: Positive | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |
  S768I: Uninformative | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 0 | 0 |  |  |  |
  S768I: Not done | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 3 | 1 |  |  |  |
  exon 20 insertions: Negative | 3 | 3 | 3 | 3 | 2 | 2 | 3 | 26 | 2 | 4 |  |  |  |
  exon 20 insertions: Positive | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |
  exon 20 insertions: Uninformative | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 0 | 0 |  |  |  |
  exon 20 insertions: Not done | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 3 | 1 |  |  |  |
  T790M: Negative | 3 | 1 | 2 | 2 | 2 | 2 | 3 | 19 | 1 | 3 |  |  |  |
  T790M: Positive | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 7 | 1 | 1 |  |  |  |
  T790M: Uninformative | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 0 | 0 |  |  |  |
  T790M: Not done | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 3 | 1 |  |  |  |

48. Secondary Outcome: Number of Participants With EGFR Mutations in Plasma in All Cohorts All Phases
Description: Number of participants with EGFR mutations in plasma in all cohorts all phases. EGFR mutation assessments in plasma included the mutations statuses of exon 19 deletion (del 19), exon 21 (L858R) and T790M.
Time Frame: Baseline
Population: as for outcome 47
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Dose-escalation: PF-06747775 25 mg QD | Phase 1 Dose-escalation: PF-06747775 50 mg QD | Phase 1 Dose-escalation: PF-06747775 150 mg QD | Phase 1 Dose-escalation: PF-06747775 275 mg QD | Phase 1 Dose-escalation: PF-06747775 300 mg QD | Phase 1 Dose-escalation: PF-06747775 450 mg QD | Phase 1 Dose-escalation: PF-06747775 600 mg QD | PF-06747775 200 mg QD Group | Phase 1 Sildenafil Sub-study: PF-06747775 300 mg QD + Sildenafil 25 mg SD | Phase 1b Cohort 2A: PF-06747775 200 mg QD + Palbociclib 100 mg QD | Phase 1 Food Effect and Rifampin DDI Sub-study: PF-06747775 + Rifampin | Phase 2 Cohort 2B: PF-06747775 + Palbociclib | Phase 2 Cohort 2B: PF-06747775 Single Agent | Phase 1b Cohort 3: PF-06747775 + Avelumab
Number analyzed (Participants) | 4 | 3 | 4 | 4 | 3 | 4 | 4 | 29 | 5 | 5 | 0 | 0 | 0 | 0
Participants
  L858R: Negative | 4 | 2 | 2 | 4 | 3 | 3 | 2 | 21 | 4 | 3 |  |  |  |
  L858R: Positive | 0 | 1 | 2 | 0 | 0 | 1 | 2 | 8 | 1 | 2 |  |  |  |
  L858R: Uninformative | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |
  T790M: Negative | 3 | 1 | 0 | 1 | 1 | 3 | 3 | 19 | 3 | 2 |  |  |  |
  T790M: Positive | 1 | 2 | 4 | 3 | 2 | 1 | 1 | 10 | 2 | 3 |  |  |  |
  T790M: Uninformative | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |
  del 19 (2235_49DEL15): Negative | 2 | 2 | 3 | 2 | 1 | 4 | 4 | 26 | 4 | 5 |  |  |  |
  del 19 (2235_49DEL15): Positive | 2 | 1 | 1 | 2 | 2 | 0 | 0 | 3 | 1 | 0 |  |  |  |
  del 19 (2235_49DEL15): Uninformative | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |
  del 19 (2236_50DEL15): Negative | 4 | 3 | 3 | 3 | 3 | 4 | 4 | 22 | 5 | 5 |  |  |  |
  del 19 (2236_50DEL15): Positive | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 6 | 0 | 0 |  |  |  |
  del 19 (2236_50DEL15): Uninformative | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 |  |  |  |
  del 19 (2237_55DELINST): Negative | 4 | 2 | 4 | 4 | 3 | 4 | 4 | 26 | 5 | 5 |  |  |  |
  del 19 (2237_55DELINST): Positive | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 |  |  |  |
  del 19 (2237_55DELINST): Uninformative | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 |  |  |  |
  del 19 (2239_48DELINSC): Negative | 4 | 3 | 4 | 4 | 3 | 4 | 4 | 29 | 5 | 4 |  |  |  |
  del 19 (2239_48DELINSC): Positive | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 |  |  |  |
  del 19 (2239_48DELINSC): Uninformative | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |
  del 19 (2240_54DEL15): Negative | 4 | 3 | 4 | 4 | 3 | 4 | 4 | 28 | 5 | 5 |  |  |  |
  del 19 (2240_54DEL15): Positive | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |
  del 19 (2240_54DEL15): Uninformative | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 |  |  |  |
  del 19 (2240_57DEL18): Negative | 4 | 2 | 4 | 4 | 3 | 3 | 4 | 27 | 5 | 5 |  |  |  |
  del 19 (2240_57DEL18): Positive | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 |  |  |  |
  del 19 (2240_57DEL18): Uninformative | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |

49. Secondary Outcome: Number of Participants With Positive Serum Anti-drug Antibody (ADA) of Avelumab in Phase 1b Cohort 3
Description: Number of participants with positive serum ADA of avelumab at pre-dose on Day 1 of Cycles 1-3 and Cycle 1 Day 15 in Phase 1b Cohort 3.
Time Frame: Pre-dose on Day 1 of Cycles 1-3 and Cycle 1 Day 15
Population: The immunogenicity analysis set included participants who had at least one ADA sample collected for avelumab.
Arm/Group | Phase 1b Cohort 3: PF-06747775 + Avelumab
Number analyzed (Participants) | 0

50. Secondary Outcome: AUCinf of PF-06747775 Following Single Dose on Lead-in Day -4 in Japan LIC RP2D Cohort, Lead-in Day -7 and Cycle 1 Day 1 in Japan LIC PK Cohort
Description: AUCinf of PF-06747775 following a 200 mg single dose on Lead-in Day -4 in Japan LIC RP2D cohort and Cycle 1 Day 1 in Japan LIC PK cohort, and following a 100 mg single dose on Lead-in Day -7 in Japan LIC PK cohort. AUCinf was defined as area under the plasma concentration versus time curve from zero to extrapolated infinite time.
Time Frame: 0 (pre-dose), 1, 2, 4, 6, 8 and 24 hours post dose on Lead-in Day -4 for Japan LIC RP2D cohort, Lead-in Day -7 and Cycle 1 Day 1 for Japan LIC PK cohort
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- Japan LIC RP2D Cohort: PF-06747775 200 mg SD => 200 mg QD: Japanese participants received a single oral dose of PF-06747775 200 mg on Day -4 in lead-in period, followed by continuous dosing of PF-06747775 200 mg QD for 21-day cycle (up to a maximum of 61 weeks).
- Japan LIC PK Cohort: PF-06747775 100 mg SD => 200 mg QD: Japanese participants received a single dose of PF-06747775 100 mg on Day -7 in lead-in period, followed by continuous dosing of PF-06747775 200 mg QD for 21-day cycle (up to a maximum of 25 weeks).
Arm/Group | Japan LIC RP2D Cohort: PF-06747775 200 mg SD => 200 mg QD | Japan LIC PK Cohort: PF-06747775 100 mg SD => 200 mg QD
Number analyzed (Participants) | 3 | 3
ng*hr/mL
  PF-06747775 200 mg SD | 13610 (39) | 16060 (4)
  PF-06747775 100 mg SD: number analyzed (Participants) | 0 | 3
  PF-06747775 100 mg SD |  | 6880 (23)

51. Secondary Outcome: Cmax of PF-06747775 Following Single Dose on Lead-in Day -4 in Japan LIC RP2D Cohort, Lead-in Day -7 and Cycle 1 Day 1 in Japan LIC PK Cohort
Description: Cmax of PF-06747775 following a 200 mg single dose on Lead-in Day -4 in Japan LIC RP2D cohort and Cycle 1 Day 1 in Japan LIC PK cohort, and following a 100 mg single dose on Lead-in Day -7 in Japan LIC PK cohort. Cmax was the maximum concentration observed from data.
Time Frame: as for outcome 50
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Japan LIC RP2D Cohort: PF-06747775 200 mg SD => 200 mg QD | Japan LIC PK Cohort: PF-06747775 100 mg SD => 200 mg QD
Number analyzed (Participants) | 3 | 3
ng/mL
  PF-06747775 200 mg SD | 3128 (22) | 2795 (36)
  PF-06747775 100 mg SD: number analyzed (Participants) | 0 | 3
  PF-06747775 100 mg SD |  | 1407 (26)

52. Secondary Outcome: Vz/F of PF-06747775 Following Single Dose on Lead-in Day -4 in Japan LIC RP2D Cohort, Lead-in Day -7 and Cycle 1 Day 1 in Japan LIC PK Cohort
Description: Vz/F of PF-06747775 following a 200 mg single dose on Lead-in Day -4 in Japan LIC RP2D cohort and Cycle 1 Day 1 in Japan LIC PK cohort, and following a 100 mg single dose on Lead-in Day -7 in Japan LIC PK cohort. Vz/F was defined as apparent volume of distribution. Vz/F was calculated as: Vz/F = dose / (AUCinf * kel). kel was defined as terminal phase rate constant and calculated by a linear regression of the log-linear concentration-time curve. AUCinf was area under the plasma concentration versus time curve (AUC) from zero to extrapolated infinite time.
Time Frame: as for outcome 50
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Japan LIC RP2D Cohort: PF-06747775 200 mg SD => 200 mg QD | Japan LIC PK Cohort: PF-06747775 100 mg SD => 200 mg QD
Number analyzed (Participants) | 3 | 3
L
  PF-06747775 200 mg SD | 90.94 (91) | 96.23 (30)
  PF-06747775 100 mg SD: number analyzed (Participants) | 0 | 3
  PF-06747775 100 mg SD |  | 108.2 (30)

53. Secondary Outcome: t1/2 of PF-06747775 Following Single Dose on Lead-in Day -4 in Japan LIC RP2D Cohort, Lead-in Day -7 and Cycle 1 Day 1 in Japan LIC PK Cohort
Description: t1/2 of PF-06747775 following a 200 mg single dose on Lead-in Day -4 in Japan LIC RP2D cohort and Cycle 1 Day 1 in Japan LIC PK cohort, and following a 100 mg single dose on Lead-in Day -7 in Japan LIC PK cohort. t1/2 was defined as the time measured for the plasma concentration to decrease by one half.
Time Frame: as for outcome 50
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: hrs
Arm/Group | Japan LIC RP2D Cohort: PF-06747775 200 mg SD => 200 mg QD | Japan LIC PK Cohort: PF-06747775 100 mg SD => 200 mg QD
Number analyzed (Participants) | 3 | 3
hrs
  PF-06747775 200 mg SD | 4.527 (1.662) | 5.563 (1.981)
  PF-06747775 100 mg SD: number analyzed (Participants) | 0 | 3
  PF-06747775 100 mg SD |  | 5.317 (1.596)

54. Secondary Outcome: AUCtau of PF-06747775 Following Multiple Doses in Japan LIC RP2D and PK Cohorts
Description: AUCtau of PF-06747775 following multiple doses on Cycle 1 Day 11 in Japan LIC RP2D cohort and Cycle 1 Day 15 in Japan LIC PK cohort. AUCtau was defined as area under the plasma concentration-time profile from time zero to tau, the dosing interval, where tau = 24 hours. AUCtau was calculated using Linear/Log trapezoidal method.
Time Frame: 0 (pre-dose), 1, 2, 4, 6, 8 and 24 hours post dose on Cycle 1 Day 11 (Japan LIC RP2D cohort) and Day 15 (Japan LIC PK cohort)
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Japan LIC RP2D Cohort: PF-06747775 200 mg SD => 200 mg QD | Japan LIC PK Cohort: PF-06747775 100 mg SD => 200 mg QD
Number analyzed (Participants) | 3 | 3
ng*hr/mL | 17680 (35) | 23300 (32)

55. Secondary Outcome: Ctrough of PF-06747775 Following Multiple Doses in Japan LIC RP2D and PK Cohorts
Description: Ctrough of PF-06747775 following multiple doses on Cycle 1 Day 11 in Japan LIC RP2D cohort and Cycle 1 Day 15 in Japan LIC PK cohort. Ctrough was defined as pre-dose concentration during multiple dosing and observed directly from data.
Time Frame: Pre-dose on Cycle 1 Day 11 (Japan LIC RP2D cohort) and Day 15 (Japan LIC PK cohort)
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Japan LIC RP2D Cohort: PF-06747775 200 mg SD => 200 mg QD | Japan LIC PK Cohort: PF-06747775 100 mg SD => 200 mg QD
Number analyzed (Participants) | 3 | 3
ng/mL | 48.91 (14) | 79.75 (91)

56. Secondary Outcome: Rac of PF-06747775 Following Multiple Doses in Japan LIC RP2D and PK Cohorts
Description: Rac of PF-06747775 following multiple doses on Cycle 1 Day 11 in Japan LIC RP2D cohort and Cycle 1 Day 15 in Japan LIC PK cohort. Rac was calculated as: Rac = (steady state AUCtau) / (single dose AUC24). AUC24 was defined as area under the plasma concentration-time curve from time 0 to 24 hours following single dose. AUCtau was defined as area under the plasma concentration-time profile from time zero to tau, the dosing interval, where tau = 24 hours.
Time Frame: 0 (pre-dose), 1, 2, 4, 6, 8 and 24 hours post dose on Lead-in Day -4, Cycle 1 Day 11 for Japan LIC RP2D cohort, Cycle 1 Days 1 and 15 for Japan LIC PK cohort
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Japan LIC RP2D Cohort: PF-06747775 200 mg SD => 200 mg QD | Japan LIC PK Cohort: PF-06747775 100 mg SD => 200 mg QD
Number analyzed (Participants) | 3 | 3
Ratio | 1.322 (50) | 1.766 (22)

57. Secondary Outcome: Rss of PF-06747775 Following Multiple Doses in Japan LIC RP2D and PK Cohorts
Description: Rss of PF-06747775 following multiple doses on Cycle 1 Day 11 in Japan RP2D cohort and Cycle 1 Day 15 in Japan PK cohort. Rss was calculated as: Rss = (steady state AUCtau) / (single dose AUCinf). AUCtau was defined as area under the plasma concentration-time profile from time zero to tau, the dosing interval, where tau = 24 hours. AUCinf was area under the plasma concentration versus time curve (AUC) from zero to extrapolated infinite time.
Time Frame: as for outcome 56
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Japan LIC RP2D Cohort: PF-06747775 200 mg SD => 200 mg QD | Japan LIC PK Cohort: PF-06747775 100 mg SD => 200 mg QD
Number analyzed (Participants) | 3 | 3
Ratio | 1.298 (49) | 1.689 (25)

58. Secondary Outcome: CL/F of PF-06747775 Following Single and Multiple Doses in Japan LIC RP2D and PK Cohorts
Description: CL/F of PF-06747775 following single dose on Lead-in Day -4 in Japan LIC RP2D cohort, Lead-in Day -7 and Cycle 1 Day 1 in Japan LIC PK cohort, and following multiple doses on Cycle 1 Day 11 in Japan LIC RP2D cohort and on Cycle 1 Day 15 in Japan LIC PK cohort. CL/F was calculated as: CL/F = dose/AUCinf for single dose or dose/AUCtau for multiple doses. AUCtau was defined as area under the plasma concentration-time profile from time zero to tau, the dosing interval, where tau = 24 hours. AUCinf was area under the plasma concentration versus time curve (AUC) from zero to extrapolated infinite time.
Time Frame: 0 (pre-dose), 1, 2, 4, 6, 8 and 24 hours post dose on Lead-in Day -4, Cycle 1 Day 11 for Japan LIC RP2D cohort, Lead-in Day-7, Days 1 and 15 for Japan LIC PK cohort
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Japan LIC RP2D Cohort: PF-06747775 200 mg SD => 200 mg QD | Japan LIC PK Cohort: PF-06747775 100 mg SD => 200 mg QD
Number analyzed (Participants) | 3 | 3
L/hr
  PF-06747775 200 mg SD | 14.64 (40) | 12.46 (4)
  PF-06747775 100 mg SD: number analyzed (Participants) | 0 | 3
  PF-06747775 100 mg SD |  | 14.57 (24)
  PF-06747775 200 mg QD | 11.32 (35) | 8.594 (32)

ADVERSE EVENTS:
Time Frame: Baseline up to 28 days after last dose of study drug (up to a maximum of 199 weeks).
Description: The same event may appear as both an AE and an SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another participant, or 1 participant may have experienced both a serious and non-serious event during the study. Total number at risk below refers to the number of participants evaluable for SAEs or AEs.
Arm/Group | Phase 1 Dose-escalation: PF-06747775 25 mg QD | Phase 1 Dose-escalation: PF-06747775 50 mg QD | Phase 1 Dose-escalation: PF-06747775 150 mg QD | Phase 1 Dose-escalation: PF-06747775 275 mg QD | Phase 1 Dose-escalation: PF-06747775 300 mg QD | Phase 1 Dose-escalation: PF-06747775 450 mg QD | Phase 1 Dose-escalation: PF-06747775 600 mg QD | PF-06747775 200 mg QD Group | Phase 1 Sildenafil Sub-study: PF-06747775 300 mg QD + Sildenafil 25 mg SD | Phase 1b Cohort 2A: PF-06747775 200 mg QD + Palbociclib 100 mg QD | Phase 1 Food Effect and Rifampin DDI Sub-study: PF-06747775 + Rifampin | Phase 2 Cohort 2B: PF-06747775 + Palbociclib | Phase 2 Cohort 2B: PF-06747775 Single Agent | Phase 1b Cohort 3: PF-06747775 + Avelumab
All-Cause Mortality (participants affected / at risk) | 0/4 | 1/3 | 0/4 | 0/4 | 0/3 | 1/4 | 1/4 | 0/29 | 0/5 | 0/5 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 2/4 | 1/3 | 3/4 | 3/4 | 0/3 | 3/4 | 2/4 | 3/29 | 0/5 | 1/5 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 4/4 | 4/4 | 3/3 | 4/4 | 4/4 | 29/29 | 5/5 | 5/5 | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 Dose-escalation: PF-06747775 25 mg QD (N=4) | Phase 1 Dose-escalation: PF-06747775 50 mg QD (N=3) | Phase 1 Dose-escalation: PF-06747775 150 mg QD (N=4) | Phase 1 Dose-escalation: PF-06747775 275 mg QD (N=4) | Phase 1 Dose-escalation: PF-06747775 300 mg QD (N=3) | Phase 1 Dose-escalation: PF-06747775 450 mg QD (N=4) | Phase 1 Dose-escalation: PF-06747775 600 mg QD (N=4) | PF-06747775 200 mg QD Group (N=29) | Phase 1 Sildenafil Sub-study: PF-06747775 300 mg QD + Sildenafil 25 mg SD (N=5) | Phase 1b Cohort 2A: PF-06747775 200 mg QD + Palbociclib 100 mg QD (N=5) | Phase 1 Food Effect and Rifampin DDI Sub-study: PF-06747775 + Rifampin (N=0) | Phase 2 Cohort 2B: PF-06747775 + Palbociclib (N=0) | Phase 2 Cohort 2B: PF-06747775 Single Agent (N=0) | Phase 1b Cohort 3: PF-06747775 + Avelumab (N=0)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Intracardiac thrombus (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 1 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 Dose-escalation: PF-06747775 25 mg QD (N=4) | Phase 1 Dose-escalation: PF-06747775 50 mg QD (N=3) | Phase 1 Dose-escalation: PF-06747775 150 mg QD (N=4) | Phase 1 Dose-escalation: PF-06747775 275 mg QD (N=4) | Phase 1 Dose-escalation: PF-06747775 300 mg QD (N=3) | Phase 1 Dose-escalation: PF-06747775 450 mg QD (N=4) | Phase 1 Dose-escalation: PF-06747775 600 mg QD (N=4) | PF-06747775 200 mg QD Group (N=29) | Phase 1 Sildenafil Sub-study: PF-06747775 300 mg QD + Sildenafil 25 mg SD (N=5) | Phase 1b Cohort 2A: PF-06747775 200 mg QD + Palbociclib 100 mg QD (N=5) | Phase 1 Food Effect and Rifampin DDI Sub-study: PF-06747775 + Rifampin (N=0) | Phase 2 Cohort 2B: PF-06747775 + Palbociclib (N=0) | Phase 2 Cohort 2B: PF-06747775 Single Agent (N=0) | Phase 1b Cohort 3: PF-06747775 + Avelumab (N=0)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 4 | 0 | 1 | 1 | 4 | 2 | 2 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bundle branch block right (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Congestive cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctival oedema (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Corneal erosion (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Erythema of eyelid (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eyelid rash (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eyelids pruritus (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Growth of eyelashes (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Macular degeneration (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pterygium (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Trichomegaly (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vitreous haemorrhage (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Anal inflammation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 3 | 2 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 4 | 3 | 4 | 4 | 20 | 4 | 5 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 3 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 1 | 3 | 0 | 1 | 1 | 5 | 1 | 2 | 0 | 0 | 0 | 0
Oesophageal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 3 | 2 | 1 | 16 | 2 | 3 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 5 | 0 | 1 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 3 | 2 | 1 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 2 | 1 | 0 | 2 | 2 | 5 | 2 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Anal fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 4 | 0 | 1 | 0 | 0 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Helicobacter gastritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Onychomycosis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 1 | 1 | 2 | 3 | 2 | 3 | 2 | 23 | 4 | 4 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 4 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tinea cruris (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 7 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 4 | 0 | 1 | 0 | 0 | 0 | 0
Blood albumin decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood calcium decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 2 | 1 | 1 | 2 | 14 | 2 | 2 | 0 | 0 | 0 | 0
Blood sodium decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood urea increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Creatinine renal clearance decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 3 | 0 | 0 | 0 | 0
Oxygen saturation decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 3 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 3 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 2 | 2 | 1 | 2 | 1 | 4 | 2 | 2 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 2 | 1 | 1 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 5 | 3 | 1 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Facial paralysis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 3 | 1 | 0 | 0 | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 3 | 0 | 2 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Azotaemia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Prostatic obstruction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vulvovaginal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal rash (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 2 | 1 | 5 | 0 | 0 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0 | 0 | 3 | 1 | 4 | 2 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 0 | 1 | 1 | 2 | 3 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3 | 3 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 0 | 1 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 1 | 3 | 1 | 9 | 3 | 2 | 0 | 0 | 0 | 0
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 3 | 1 | 1 | 0 | 7 | 1 | 1 | 0 | 0 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 2 | 3 | 1 | 15 | 2 | 2 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 4 | 1 | 3 | 1 | 14 | 1 | 2 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 3 | 2 | 2 | 1 | 8 | 2 | 2 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 3 | 4 | 3 | 4 | 2 | 13 | 4 | 3 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 2 | 7 | 0 | 0 | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2016-12-19): https://cdn.clinicaltrials.gov/large-docs/33/NCT02349633/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-05): https://cdn.clinicaltrials.gov/large-docs/33/NCT02349633/SAP_001.pdf